CLINICAL TRIAL: NCT03446573
Title: A Phase III, Randomized, Multicenter, Parallel-group, Non-inferiority Study Evaluating the Efficacy, Safety, and Tolerability of Switching to Dolutegravir Plus Lamivudine in HIV-1 Infected Adults Who Are Virologically Suppressed
Brief Title: Switch Study to Evaluate Dolutegravir Plus Lamivudine in Virologically Suppressed Human Immunodeficiency Virus Type 1 Positive Adults (TANGO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 204862; 2015-004401-17 (EudraCT Number)
Record Dates: First submitted 2018-01-05; First posted 2018-02-27 (Actual); Results first posted 2020-06-02 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: HIV Infections
Keywords: Switch study; Non-inferiority; Human immunodeficiency virus type 1; Tenofovir alafenamide; Dolutegravir; Lamivudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: This is a randomized study with parallel group assignment where participants will be randomized into one of the two treatment groups. Participants randomized to DTG + 3TC will receive DTG + 3TC up to Week 200. Participants randomized to TBR will continue to take their current regimen up to Week 148, at which time and if HIV-1 RNA <50 c/mL at Week 144, these participants will switch to DTG + 3TC up to Week 200. Randomization will be stratified by Baseline third agent class (protease inhibitor [PI], integrase inhibitor [INI], or non-nucleoside reverse transcriptase inhibitor [NNRTI]).
Masking Description: This will be an open-label study and therefore no blinding is required. No summaries of the study data according to actual randomized treatment groups will be available to sponsor staff prior to the planned Week 24 preliminary analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DTG + 3TC 50 mg/300 mg (Experimental): Participants will receive a single tablet of a two-drug regimen of DTG 50 mg + 3TC 300 mg once daily from Day 1 through Week 200 (Early and Late Switch Phase).
  Interventions: Drug: DTG + 3TC
- TAF based regimen (TBR) (Active Comparator): Participants will continue their TBR from Day 1 to Week 148 (Early Switch Phase), and eligible participants will switch to DTG + 3TC once daily from Week 148 to 200 (Late Switch Phase).
  Interventions: Drug: TAF based regimen (TBR)

INTERVENTIONS:
Drug: DTG + 3TC — DTG+3TC is supplied as white, oval, film-coated, fixed dose combination tablet. The tablets will be available in packed high density polyethylene (HDPE) bottles with induction seals and child-resistant closures.
  Arms: DTG + 3TC 50 mg/300 mg
Drug: TAF based regimen (TBR) — Participants will continue to receive their TBR.
  Arms: TAF based regimen (TBR)

SUMMARY:
The aim of the study is to establish if human immunodeficiency virus type 1 (HIV-1) infected adult participants with current virologic suppression on a >=3-drug tenofovir alafenamide (TAF) based regimen (TBR) remain suppressed upon switching to a two-drug regimen of dolutegravir (DTG) 50 milligram (mg) + lamivudine (3TC) 300 mg. This study will also provide important information regarding the safety and participant satisfaction with this two-drug regimen. The primary objective of this trial is to demonstrate the non-inferior antiviral activity of switching to DTG + 3TC once daily compared to continuation of TBR over 48 weeks in HIV-1 infected, antiretroviral therapy (ART)-experienced, virologically suppressed participants. This study also will characterize the long-term antiviral activity, tolerability and safety of DTG + 3TC compared to TBR through Week 144 and characterize the long-term antiviral activity, tolerability and safety of DTG + 3TC through Week 200.

This will be a 200-week, Phase III, randomized, open-label, active-controlled, multicenter, parallel- group study. The study will include a screening phase (up to 28 days), a randomized early switch phase (Day 1 up to Week 148), a randomized late switch phase (Week 148 up to Week 200), and a continuation phase (post Week 200). HIV-1 infected adults on stable TBR will be randomized 1:1 to switch to DTG + 3TC once daily for up to 200 weeks, or to continue their TBR for 148 weeks, at which time and if HIV-1 ribonucleic acid (RNA) <50 copies per milliliter (c/mL) at Week 144, these participants will switch to DTG + 3TC up to Week 200.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be able to understand and comply with protocol requirements, instructions, and restrictions;
* Participant must be likely to complete the study as planned;
* Participant must be considered an appropriate candidate for participation in an investigative clinical trial with medication (example no active substance abuse, acute major organ disease, or planned long-term work assignments out of the country).
* Aged 18 years or older (or older where required by local regulatory agencies), at the time of signing the informed consent.
* HIV-1 infected men or women.
* Documented evidence of at least two plasma HIV-1 RNA measurements <50 c/mL in the 12 months prior to Screening: one within the 6 to 12 month window, and one within 6 months prior to Screening.
* Plasma HIV-1 RNA <50 c/mL at Screening.
* Must be on uninterrupted ART for at least 6 months prior to screening. Only the following regimens are allowed:

  * Participant on a TAF-based regimen for at least 6 months as the initial regimen, or
  * Participants who switched from a tenofovir disoproxil fumarate (TDF) first-regimen TAF, without any changes to the other drugs in their regimen, and have been on the TAF-based regimen for at least 3 months immediately prior to Screening i.e., the only switch made is from TDF to TAF. This switch must have occurred due to tolerability/safety, access to medications, or convenience/simplification, and must NOT have been done for suspected or established treatment failure. A switch from a PI boosted with ritonavir to the same PI boosted with cobicistat is allowed (and vice versa).
* A female participant is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin [hCG] test at screen and a negative urine hCG test at randomization [a local serum hCG test at Randomization is allowed if it can be done, and results obtained, within 24 hours prior to randomization]), not lactating, and at least one of the following conditions applies:

  a. Non-reproductive potential defined as:
* Pre-menopausal females with one of the following:

  * Documented tubal ligation
  * Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion
  * Hysterectomy
  * Documented bilateral oophorectomy
* Post-menopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause [refer to laboratory reference ranges for confirmatory levels]). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

  b. Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and for at least 2 weeks after the last dose of study medication.
* The investigator is responsible for ensuring that participants understand how to properly use these methods of contraception. All participants participating in the study should be counseled on safer sexual practices including the use and benefit/risk of effective barrier methods (e.g., male condom) and on the risk of HIV transmission to an uninfected partner.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and the protocol. Eligible participants or their legal guardians must sign a written informed consent form before any protocol-specified assessments are conducted.

Participants enrolled in France must be affiliated to, or a beneficiary of, a social security category.

Exclusion Criteria:

* Women who are breastfeeding or plan to become pregnant or breastfeed during the study.
* Any evidence of an active Centers for Disease Control and Prevention (CDC) Stage 3 disease, EXCEPT cutaneous Kaposi's sarcoma not requiring systemic therapy. Historical or current CD4 cell counts less than 200 cells/millimeter (mm)^3 are NOT exclusionary.
* Participants with severe hepatic impairment (Class C) as determined by Child-Pugh classification.
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antigen antibody (anti-HBs) and HBV deoxyribonucleic acid (DNA) as follows: participants positive for HBsAg are excluded; participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded.
* Anticipated need for any hepatitis C virus (HCV) therapy during the first 48 weeks of the study, or anticipated need for HCV therapy based on interferon or for any drugs that have a potential for adverse drug-drug interactions with study treatment throughout the entire study period.
* Untreated syphilis infection (positive rapid plasma reagin [RPR] at Screening without clear documentation of treatment). Participants who are at least 7 days post completed treatment are eligible.
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia.
* Participants who in the investigator's judgment, poses a significant suicidality risk.
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
* Treatment with any of the following agents within 28 days of Screening: radiation therapy; cytotoxic chemotherapeutic agents; any systemic immune suppressant.
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of investigational product (IP).
* Use of any regimen consisting of single or dual ART.
* Any evidence of major nucleoside reverse transcriptase inhibitor (NRTI) mutation or presence of any major INSTI resistance-associated mutation in any available prior resistance genotype assay test result, if known, must be provided to ViiV after screening and before randomization for review by ViiV Virology.
* Any verified Grade 4 laboratory abnormality.
* Alanine aminotransferase (ALT) >=5 times (*) the upper limit of normal (ULN) or ALT >=3 * ULN and bilirubin >=1.5 * ULN (with >35 percent [%] direct bilirubin).
* Creatinine clearance of <50 milliliter (mL)/minute/1.73 meter^2 via Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) method.
* Within the 6 to 12 month window prior to Screening and after confirmed suppression to <50 c/mL, any plasma HIV-1 RNA measurement >200 c/mL.
* Within the 6 to 12 month window prior to Screening and after confirmed suppression to <50 c/mL, 2 or more plasma HIV-1 RNA measurements >=50 c/mL.
* Within 6 months prior to Screening and after confirmed suppression to <50 c/mL on current ART regimen, any plasma HIV-1 RNA measurement >=50 c/mL.
* Any drug holiday during the 6 months prior to Screening, except for brief periods (less than 1 month) where all ART was stopped due to tolerability and/or safety concerns.
* Any history of switch to another regimen, defined as change of a single drug or multiple drugs simultaneously, due to virologic failure to therapy (defined as a confirmed plasma HIV-1 RNA ≥400 c/mL.
* Participants enrolled in France (or in other countries as required by local regulations or Ethics Committee/Institutional Review Board [IRB]) who:

  * Participated in any study using an investigational drug or vaccine during the previous 60 days or 5 half-lives, or twice the duration of the biological effect of the experimental drug or vaccine, whichever is longer, prior to screening for the study, or
  * Participate simultaneously in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2022-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (107):
- United States (47):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Rialto, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Leandro, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Beach, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Berkley, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lynchburg, Virginia
- Australia (9):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Darlinghurst, Sydney, New South Wales
  - GSK Investigational Site, Surry Hills, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Fortitude Valley, Queensland
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Fitzroy North, Victoria
  - GSK Investigational Site, Prahran, Victoria
- Belgium (3):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
- Canada (3):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (5):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Tourcoing
- Germany (7):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, München
- Japan (3):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Rotterdam, Netherlands
- Spain (22):
  - GSK Investigational Site, Vigo, Galicia
  - GSK Investigational Site, Alcalá de Henares
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cartagena (Murcia)
  - GSK Investigational Site, Elche
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Granollers (Barcelona)
  - GSK Investigational Site, Huelva
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vilajoyosa
  - GSK Investigational Site, Zaragoza
- United Kingdom (7):
  - GSK Investigational Site, Birmingham, West Midlands
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Brighton
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Crumpsall, Manchester
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on ViiV's data sharing criteria can be found at: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/

REFERENCES:
- [Background] van Wyk J, Ajana F, Bisshop F, De Wit S, Osiyemi O, Portilla Sogorb J, Routy JP, Wyen C, Ait-Khaled M, Nascimento MC, Pappa KA, Wang R, Wright J, Tenorio AR, Wynne B, Aboud M, Gartland MJ, Smith KY. Efficacy and Safety of Switching to Dolutegravir/Lamivudine Fixed-Dose 2-Drug Regimen vs Continuing a Tenofovir Alafenamide-Based 3- or 4-Drug Regimen for Maintenance of Virologic Suppression in Adults Living With Human Immunodeficiency Virus Type 1: Phase 3, Randomized, Noninferiority TANGO Study. Clin Infect Dis. 2020 Nov 5;71(8):1920-1929. doi: 10.1093/cid/ciz1243. PMID 31905383
- [Derived] Scholten S, Cahn P, Portilla J, Bisshop F, Hodder S, Ruane P, Kaplan R, Wynne BR, Man CY, Grove R, Wang R, Jones B, Ait-Khaled M, Kisare M, Okoli C. Dolutegravir/Lamivudine Efficacy and Safety Outcomes in People With HIV-1 With or Without Historical Resistance Results at Screening: 48-Week Pooled Analysis. Open Forum Infect Dis. 2024 Jul 1;11(7):ofae365. doi: 10.1093/ofid/ofae365. eCollection 2024 Jul. PMID 39015350
- [Derived] Ait-Khaled M, Oyee J, Ooi AYR, Wynne B, Maldonado A, Jones B, Wang T. Efficacy and Safety of Switching to Dolutegravir/Lamivudine Versus Continuing a Tenofovir Alafenamide-Based Regimen in Virologically Suppressed Adults With Human Immunodeficiency Virus Type 1: Subgroup Analysis of Participants With Elvitegravir as Baseline Third Agent From the TANGO Study. Open Forum Infect Dis. 2024 May 2;11(5):ofae227. doi: 10.1093/ofid/ofae227. eCollection 2024 May. PMID 38737429
- [Derived] Chandasana H, Singh R, Adkison K, Ait-Khaled M, Pene Dumitrescu T. Population pharmacokinetic modeling of dolutegravir/lamivudine to support a once-daily fixed-dose combination regimen in virologically suppressed adults living with HIV-1. Antimicrob Agents Chemother. 2024 May 2;68(5):e0150423. doi: 10.1128/aac.01504-23. Epub 2024 Apr 8. PMID 38587380
- [Derived] Walmsley S, Smith DE, Gorgolas M, Cahn PE, Lutz T, Lacombe K, Kumar PN, Wynne B, Grove R, Bontempo G, Moodley R, Okoli C, Kisare M, Jones B, Clark A, Ait-Khaled M. Efficacy and safety of switching to dolutegravir/lamivudine in virologically suppressed people with HIV-1 aged >/= 50 years: week 48 pooled results from the TANGO and SALSA studies. AIDS Res Ther. 2024 Mar 21;21(1):17. doi: 10.1186/s12981-024-00604-9. PMID 38515183
- [Derived] Wang R, Underwood M, Llibre JM, Bernal Morell E, Brinson C, Sanz Moreno J, Scholten S, Moore R, Saggu P, Oyee J, Moodley R, Wynne B, Kisare M, Jones B, Ait-Khaled M. Very-Low-Level Viremia, Inflammatory Biomarkers, and Associated Baseline Variables: Three-Year Results of the Randomized TANGO Study. Open Forum Infect Dis. 2023 Dec 9;11(1):ofad626. doi: 10.1093/ofid/ofad626. eCollection 2024 Jan. PMID 38213637
- [Derived] Batterham RL, Espinosa N, Katlama C, McKellar M, Scholten S, Smith DE, Ait-Khaled M, George N, Wright J, Gordon LA, Moodley R, Wynne B, van Wyk J. Cardiometabolic Parameters 3 Years After Switch to Dolutegravir/Lamivudine vs Maintenance of Tenofovir Alafenamide-Based Regimens. Open Forum Infect Dis. 2023 Jul 12;10(7):ofad359. doi: 10.1093/ofid/ofad359. eCollection 2023 Jul. PMID 37520420
- [Derived] Wang R, Wright J, Saggu P, Ait-Khaled M, Moodley R, Parry CM, Lutz T, Podzamczer D, Moore R, Gorgolas Hernandez-Mora M, Kinder C, Wynne B, van Wyk J, Underwood M. Assessing the Virologic Impact of Archived Resistance in the Dolutegravir/Lamivudine 2-Drug Regimen HIV-1 Switch Study TANGO through Week 144. Viruses. 2023 Jun 11;15(6):1350. doi: 10.3390/v15061350. PMID 37376649
- [Derived] Osiyemi O, De Wit S, Ajana F, Bisshop F, Portilla J, Routy JP, Wyen C, Ait-Khaled M, Leone P, Pappa KA, Wang R, Wright J, George N, Wynne B, Aboud M, van Wyk J, Smith KY. Efficacy and Safety of Switching to Dolutegravir/Lamivudine Versus Continuing a Tenofovir Alafenamide-Based 3- or 4-Drug Regimen for Maintenance of Virologic Suppression in Adults Living With Human Immunodeficiency Virus Type 1: Results Through Week 144 From the Phase 3, Noninferiority TANGO Randomized Trial. Clin Infect Dis. 2022 Sep 29;75(6):975-986. doi: 10.1093/cid/ciac036. PMID 35079789
- [Derived] van Wyk J, Ait-Khaled M, Santos J, Scholten S, Wohlfeiler M, Ajana F, Jones B, Nascimento MC, Tenorio AR, Smith DE, Wright J, Wynne B. Brief Report: Improvement in Metabolic Health Parameters at Week 48 After Switching From a Tenofovir Alafenamide-Based 3- or 4-Drug Regimen to the 2-Drug Regimen of Dolutegravir/Lamivudine: The TANGO Study. J Acquir Immune Defic Syndr. 2021 Jun 1;87(2):794-800. doi: 10.1097/QAI.0000000000002655. PMID 33587500

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-inferiority study evaluated antiviral activity of switching to dolutegravir (DTG) + lamivudine (3TC) fixed dose combination (FDC) once daily compared to continuation of a Tenofovir alafenamide (TAF)-based regimen (TBR) over 148 weeks in virologically suppressed participants with human immunodeficiency type 1 infection. At week 148 all participants received DTG + 3TC FDC until week 196.
Pre-assignment Details: A total of 743 participants were randomized to receive treatment. Two participants in the DTG+3TC group were randomized but not treated. A total of 741 participants received at least one dose of study treatment either DTG + 3TC or TBR creating the intent to treat-exposed (ITT-E) Population.
Groups:
- DTG+3TC FDC: Participants who were on a stable TBR and who had an HIV-1 ribonucleic acid (RNA) less than (<)50 copies per millilter (c/mL) at the time of screening, received fixed dose combination of DTG 50 milligrams (mg) + 3TC 300 mg in early switch phase (Day 1 to Week 148) and continued to receive DTG/3TC FDC in late switch phase (Week 148 to Week 196).
- TAF-based Regimen: Participants who were on a stable TBR and had an HIV-1 RNA<50 c/mL at the time of screening received TBR up to Week 148 in early switch phase, these participants were switched to DTG/3TC FDC in late switch phase (Week 148 to Week 196). One participant randomized to this arm received TDF rather than TAF-and was presented within the "TAF-based regimen" arm (early switch phase) for efficacy because the efficacy of TAF and TDF are comparable. However, the participant was presented separately under "TDF-based regimen"arm (early switch phase) for Safety because the safety profiles of TDF and TAF differ.
Period: Early Switch Phase (Day 1 to Week 148)
Arm/Group | DTG+3TC FDC | TAF-based Regimen
Started (Randomised) | 371 | 372
ITT-E Population | 369 | 372
Completed | 319 | 299
Not Completed | 52 | 73
Not completed — Adverse Event | 23 | 7
Not completed — Lack of Efficacy | 0 | 6
Not completed — Protocol Violation | 5 | 6
Not completed — Lost to Follow-up | 4 | 10
Not completed — Physician Decision | 2 | 11
Not completed — Withdrawal by Subject | 16 | 33
Not completed — Randomized, but did not receive treatment | 2 | 0
Period: Late Switch Phase (Week 148 to Week 196)
Arm/Group | DTG+3TC FDC | TAF-based Regimen
Started | 319 | 298 (One participant was not switched to DTG+ 3TC FDC due to being lost to follow up post Week 148 visit, hence did not enter in the late switch phase)
Completed | 307 | 274
Not Completed | 12 | 24
Not completed — Adverse Event | 2 | 9
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 5 | 6
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 4 | 6

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics data are reported for participants in the ITT-E Population
Groups:
- Total: Total of all reporting groups
Arm/Group | DTG+3TC FDC | TAF-based Regimen | Total
Number analyzed (Participants) | 369 | 372 | 741
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.6 (10.76) | 40.9 (11.54) | 40.8 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 33 | 58
  Male | 344 | 339 | 683
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 8 | 15
  Asian-Central/South Asian Heritage (H) | 3 | 4 | 7
  Asian-Japanese H/East Asian H/South East Asian H | 10 | 9 | 19
  Black or African American | 50 | 58 | 108
  Native Hawaiian or other Pacific Islander | 1 | 3 | 4
  White-Arabic/North African (NA) H | 5 | 2 | 7
  White-Arabic/NA H and white/caucasia/European H | 0 | 1 | 1
  White-White/caucasian/European H | 292 | 286 | 578
  Asian and White | 0 | 1 | 1
  Black or African American and White | 1 | 0 | 1
Cluster of differentiation 4 plus (CD4+) cell count [Median (Inter-Quartile Range); unit: Cells per cubic millimeter (cells/mm^3)] — Blood samples were collected to evaluate Baseline CD4+ cell count using flow cytometry. Median along with first and third quartiles are presented for Baseline CD4+ count.
  Cells per cubic millimeter (cells/mm^3) | 682.0 [492.0 to 862.0] | 720.0 [531.5 to 901.5] | 688.0 [514.0 to 885.0]
Baseline third agents [Count of Participants; unit: Participants] — Baseline third agents including non-nucleoside reverse transcriptase inhibitors (NNRTI), integrase strand transfer inhibitors (INSTI) and protease inhibitors (PI) based on the antiretroviral medications taken at Baseline.
  Participants
    NNRTI | 51 | 48 | 99
    INSTI | 289 | 296 | 585
    PI | 29 | 28 | 57
HIV infection by Centers for Disease Control and Prevention (CDC) classification [Count of Participants; unit: Participants] — CDC classification for human immunodeficiency (HIV) were: Stage 1: No acquired immuno deficiency syndrome (AIDS) defining condition and CD4+ T-lymphocyte count: >=500 cells per microliter (cells/mcL); Stage 2: No AIDS-defining condition and CD4 200-499; Stage 3: Documentation of an AIDS- defining condition or CD4 < 200cells/mcL .
  Participants
    HIV infection Stage 1 | 255 | 259 | 514
    HIV infection Stage 2 | 94 | 94 | 188
    HIV infection Stage 3 | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Virologic Failure Endpoint as Per Food and Drug Administration (FDA) Snapshot Category at Week 48
Description: Percentage of participants with virologic failure (plasma HIV-1 RNA >=50 c/mL) was evaluated using FDA snapshot algorithm at Week 48. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant antiretroviral therapy (ART) prior to the visit of interest. Intent-to-treat exposed (ITT-E) Population comprises of all randomized participants who received at least one dose of study treatment either DTG + 3TC or TBR. Participants were assessed according to the treatment to which the participant was randomized. Any participant receiving a treatment randomization number was considered to be randomized.
Time Frame: Week 48
Population: ITT-E Population. One participant randomized to TBR but received TDF-based regimen and was presented within the "TBR (TAF-based regimen) arm" as efficacy of TAF and TDF are comparable.
Measure: Number; unit: Percentage of participants
Groups:
- DTG+3TC FDC (Early Switch): Participants who were on a stable TBR and who had an HIV-1 ribonucleic acid (RNA) <50 copies per millilter (c/mL) at the time of screening, received fixed dose combination of DTG 50 milligrams (mg) + 3TC 300 mg once daily up to 148 weeks during early switch phase.
- TAF Based Regimen (Early Switch): Participants who were on a stable TBR and who had an HIV-1 RNA<50 c/mL at the time of screening, received TBR up to 148 weeks during early switch phase. One participant randomized to the TAF-based regimen arm received TDF rather than TAF-and was presented within the "TAF-based regimen" arm for efficacy because the efficacy of TAF and TDF are comparable. However, the participant was presented separately under "TDF-based regimen" for Safety because the safety profiles of TDF and TAF differ.
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 372
Percentage of participants | 0.3 | 0.5
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Non-Inferiority — Non-inferiority of switching to DTG + 3TC compared to continuation of TBR (as per FDA snapshot algorithm) was to be concluded if the upper bound of a two-sided 95% confidence interval (CI) for the difference in virologic failure rates between the two treatment arms was smaller than 4%; Adjusted difference in proportion (ADP) = -0.3, 95% CI 2-sided [-1.2 to 0.7] — ADP was based on Cochran-Mantel Haenszel stratified analysis adjusting for Baseline stratification factor:Baseline third agent (protease inhibitor [PI], non-nucleoside reverse transcriptase inhibitor [NNRTI], and integrase inhibitor [INI])

2. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL as Per Snapshot Algorithm at Week 48
Description: Percentage of participants with plasma HIV-1 RNA <50 c/mL (virologic success) was evaluated using FDA snapshot algorithm at Week 48 to demonstrate the non-inferior antiviral activity of switching to DTG +3TC once daily compared to continuation of TBR over 48 weeks. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant ART prior to the visit of interest.
Time Frame: Week 48
Population: ITT-E Population. Only those participants with data available at specified time points has been analyzed. One participant randomized to TBR but received TDF-based regimen and was presented within the "TBR (TAF-based regimen) arm" as efficacy of TAF and TDF are comparable.
Measure: Number; unit: Percentage of participants
Groups:
- TAF Based Regimen (Early Switch): Participants who were on a stable TBR and who had an HIV-1 RNA<50 c/mL at the time of screening, were continued to receive TBR up to 148 weeks during early switch phase. One participant randomized to the TAF-based regimen arm received TDF rather than TAF-and was presented within the "TAF-based regimen" arm for efficacy because the efficacy of TAF and TDF are comparable. However, the participant was presented separately under "TDF-based regimen" for Safety because the safety profiles of TDF and TAF differ.
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 344 | 346
Percentage of participants | 93.2 | 93.0
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Non-Inferiority — Non-inferiority of switching to DTG + 3TC compared to continuation of TBR (as per FDA snapshot algorithm) was to be concluded when the lower bound of a 2-sided 95% confidence interval for the difference in success rates between the two treatment arms was greater than -8%; Adjusted difference in proportion = 0.2, 95% CI 2-sided [-3.4 to 3.9] — ADP was based on Cochran-Mantel Haenszel stratified analysis adjusting for Baseline stratification factor: Baseline third agent (PI, NNRTI, and INSTI)

3. Secondary Outcome: Percentage of Participants With Virologic Failure Endpoint as Per FDA Snapshot Category at Week 24
Description: Percentage of participants with plasma HIV-1 RNA >=50 c/mL was evaluated using FDA snapshot algorithm at Week 24. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant ART prior to the visit of interest.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 372
Percentage of participants | 0.3 | 0.8

4. Secondary Outcome: Percentage of Participants With Virologic Failure Endpoint as Per FDA Snapshot Category at Weeks 96, 144
Description: Percentage of participants with plasma HIV-1 RNA >=50 c/mL was evaluated using FDA snapshot algorithm at Weeks 96 and 144.
Time Frame: Weeks 96 and 144
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- TAF-based Regimen (Early Switch): Participants who were on a stable TBR and who had an HIV-1 RNA<50 c/mL at the time of screening, were continued to receive TBR up to 148 weeks during early switch phase. One participant randomized to the TAF-based regimen arm received TDF rather than TAF-and was presented within the "TAF-based regimen" arm for efficacy because the efficacy of TAF and TDF are comparable. However, the participant was presented separately under "TDF-based regimen" for Safety because the safety profiles of TDF and TAF differ.
Arm/Group | DTG+3TC FDC (Early Switch) | TAF-based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 372
Percentage of participants
  Week 96 | 0.3 | 1.1
  Week 144 | 0.3 | 1.3

5. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL as Per Snapshot Algorithm at Week 24
Description: Percentage of participants with plasma HIV-1 RNA <50 c/mL was evaluated using FDA snapshot algorithm at Week 24. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant ART prior to the visit of interest. Percentage values are rounded off.
Time Frame: Week 24
Population: ITT-E Population. Only those participants with data available at specified time points has been presented. One participant randomized to TBR but received TDF-based regimen and was presented within the "TBR (TAF-based regimen) arm" as efficacy of TAF and TDF are comparable.
Measure: Number; unit: Percentage of participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 350 | 358
Percentage of participants | 95 | 96

6. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL as Per Snapshot Algorithm at Weeks 96 and 144
Description: Percentage of participants with plasma HIV-1 RNA <50 c/mL was evaluated using FDA snapshot algorithm at Weeks 96 and 144.
Time Frame: Weeks 96 and 144
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF-based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 372
Percentage of participants
  Week 96 | 85.9 | 79.0
  Week 144 | 85.9 | 81.7

7. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Weeks 24 and 48
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+. It was evaluated by flow cytometry. Baseline value is defined as the latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. One participant randomized to TBR but received TDF-based regimen and was presented within the "TBR (TAF-based regimen) arm" as efficacy of TAF and TDF are comparable.
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: ITT-E Population. All 741 (369+372) participants were analyzed, however only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Median (Inter-Quartile Range); unit: Cells per cubic millimeter
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 372
Cells per cubic millimeter
  Week 24, n=351, 359: number analyzed (Participants) | 351 | 359
  Week 24, n=351, 359 | 21.0 [-68.0 to 115.0] | 6.0 [-87.0 to 99.0]
  Week 48, n=344, 345: number analyzed (Participants) | 344 | 345
  Week 48, n=344, 345 | 22.5 [-71.0 to 121.5] | 11.0 [-98.0 to 90.0]

8. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Weeks 96 and 144
Description: CD4+ cells are a type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+and evaluated by flow cytometry. Baseline value is defined as the latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. One participant randomized to TBR but received TDF-based regimen and was presented within the "TBR (TAF-based regimen) arm" as efficacy of TAF and TDF are comparable
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Median (Inter-Quartile Range); unit: Cells per cubic millimeter
Arm/Group | DTG+3TC FDC (Early Switch) | TAF-based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 372
Cells per cubic millimeter
  Week 96, n=315, 295: number analyzed (Participants) | 315 | 295
  Week 96, n=315, 295 | 61.0 [-61.0 to 179.0] | 45.0 [-80.0 to 154.0]
  Week 144, n=309, 301: number analyzed (Participants) | 309 | 301
  Week 144, n=309, 301 | 36.0 [-64.0 to 154.0] | 35.0 [-60.0 to 134.0]

9. Secondary Outcome: Change From Baseline in CD4+/CD8+ Cell Count Ratio at Weeks 24 and 48
Description: Blood samples were collected at specified time points to assess CD4+/CD8+ cell count ratio. It was assessed by flow cyclometry to evaluate the immunologic activity of switching to DTG+3TC once daily compared to continuation of TBR over 48 Weeks. Baseline (Day 1) values were the actual CD4+ cell count ratio values at pre-dose Day 1. Change from Baseline is defined as post-dose visit value minus Baseline value. One participant randomized to TBR but received TDF-based regimen and was presented within the "TBR (TAF-based regimen) arm" as efficacy of TAF and TDF are comparable .
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 372
Ratio
  Week 24, n=346, 358: number analyzed (Participants) | 346 | 358
  Week 24, n=346, 358 | 0.010 [-0.070 to 0.110] | 0.040 [-0.060 to 0.120]
  Week 48, n=342, 343: number analyzed (Participants) | 342 | 343
  Week 48, n=342, 343 | 0.030 [-0.050 to 0.110] | 0.050 [-0.050 to 0.160]

10. Secondary Outcome: Change From Baseline in CD4+/CD8+ Cell Count Ratio at Weeks 96 and 144
Description: Blood samples were collected at specified time points to assess CD4+/CD8+ cell count ratio and were evaluated by flow cyclometry to evaluate the immunologic activity of switching to DTG+3TC once daily compared to continuation of TBR over Weeks 96 and 144. Baseline (Day 1) values are the actual CD4+ cell count ratio values at pre-dose Day 1. Change from Baseline is defined as post-dose visit value minus Baseline value. One participant randomized to TBR but received TDF-based regimen and was presented within the "TBR (TAF-based regimen) arm" as efficacy of TAF and TDF are comparable
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | DTG+3TC FDC (Early Switch) | TAF-based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 372
Ratio
  Week 96, n=312, 292: number analyzed (Participants) | 312 | 292
  Week 96, n=312, 292 | 0.035 [-0.085 to 0.140] | 0.080 [-0.050 to 0.170]
  Week 144, n=307, 300: number analyzed (Participants) | 307 | 300
  Week 144, n=307, 300 | 0.060 [-0.060 to 0.200] | 0.100 [-0.020 to 0.240]

11. Secondary Outcome: Number of Participants With Disease Progression at Weeks 24 and 48
Description: HIV-associated conditions were recorded during the study and were assessed according to the 2014 CDC Classification System for HIV Infection in Adults. CDC classification for HIV were: Stage 1: No AIDS defining condition and CD4+ T-lymphocyte count: >=500 cells/mcL; Stage 2: No AIDS infection and CD4+ lymphocyte count: 200-499 cell/mcL and Stage 3:Documented AIDS defining condition or CD4+ T-lymphocye count <200 cells/mcL. Disease progression summarize participants who had HIV infection stage 3 associated conditions or death. Indicators of clinical disease progression were defined as: CDC Category Stage 1 at enrollment to Stage 3 event; CDC Category Stage 2 at enrollment to Stage 3 event; CDC Category Stage 3 at enrollment to New Stage 3 Event; CDC Category Stage 1, 2 or 3 at enrollment to Death.
Time Frame: At Weeks 24 and 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 372
Participants
  From CDC Stage 1 to CDC Stage 3 Event | 1 | 0
  From CDC Stage 2 to CDC Stage 3 Event | 0 | 0
  From CDC Stage 3 to new CDC Stage 3 Event | 0 | 0
  From CDC Stage 1, 2 or 3 to Death | 1 | 0
  No HIV-1 disease progression | 367 | 372

12. Secondary Outcome: Number of Participants With Disease Progression at Weeks 96 and 144
Description: HIV-associated conditions were recorded during the study and assessed according to the 2014 CDC Classification System for HIV Infection in Adults. CDC classification for HIV is: Stage 1: No AIDS defining condition and CD4+ T-lymphocyte count: >=500 cells/mcL; Stage 2: No AIDS infection and CD4+ lymphocyte count: 200-499 cell/mcL and Stage 3: Documented AIDS-defining condition or CD4+ T-lymphocye count <200 cells/mcL. Indicators of clinical disease progression is defined as: CDC Category Stage 1 at enrollment to Stage 3 event; CDC Category Stage 2 at enrollment to Stage 3 event; CDC Category Stage 3 at enrollment to New Stage 3 Event; CDC Category Stage 1, 2 or 3 at enrollment to Death.
Time Frame: At Weeks 96 and 144
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF-based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 372
Participants
  Week 96, From CDC Stage 1 to CDC Stage 3 Event | 2 | 0
  Week 96, From CDC Stage 2 to CDC Stage 3 Event | 0 | 0
  Week 96, From CDC Stage 3 to new CDC Stage 3 Event | 0 | 0
  Week 96, From CDC Stage 1, 2 or 3 to Death | 2 | 0
  Week 96, No HIV-1 disease progression | 365 | 372
  Week 144, From CDC Stage 1 to CDC Stage 3 Event | 2 | 0
  Week 144, From CDC Stage 2 to CDC Stage 3 Event | 0 | 1
  Week 144,From CDC Stage 3 to new CDC Stage 3 Event | 0 | 0
  Week 144, From CDC Stage 1, 2 or 3 to Death | 3 | 0
  Week 144, No HIV-1 disease progression | 364 | 371

13. Secondary Outcome: Number of Participants With Any Serious Adverse Events (SAEs) and Common (>=2%) Non-serious Adverse Events (Non-SAEs): Up to Week 48
Description: An AE is any untoward medical occurrence temporally associated with the use of a study treatment, whether or not considered related to study treatment. A SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other important medical event as per medical or scientific judgment . Safety Population included all participants who received at least one dose of study treatment either DTG + 3TC or TBR. This population was based on the treatment the participant actually received. Number of participants with any SAE and common (>=2%) non-SAEs are presented.
Time Frame: Up to Week 48
Population: Safety Population. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Participants
  Any non-SAE (>=2%) | 222 | 204
  Any SAE | 21 | 16

14. Secondary Outcome: Number of Participants Randomized to TBR Arm Receiving TDF-based Regimen With Any SAEs and Common (>=2%) Non-SAEs: Up to Week 48
Description: An AE is any untoward medical occurrence temporally associated with the use of a study treatment, whether or not considered related to study treatment. A SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other important medical event as per medical or scientific judgment . Number of TDF-based regimen participants with any SAE and common (>=2%) non-SAEs are presented.
Time Frame: Up to Week 48
Population: Safety Population. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."Data not collected post week 48 as the participant withdrew from the study.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized to TBR But Received TDF-based Regimen (Early Switch): Participant randomized to TBR arm who had HIV-1 RNA <50 c/mL at the time of screening, received TDF-based regimen instead of TAF-based regimen in error. Participant continued to receive TDF-regimen up to the Week 48 visit (participant withdrew from the study at Week 36)
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Participants
  Any non-SAE (>=2%) | 1
  Any SAE | 0

15. Secondary Outcome: Number of Participants With Any SAEs and Common (>=2%) Non-SAEs: Up to Week 148
Description: An AE is any untoward medical occurrence temporally associated with the use of a study treatment, whether or not considered related to study treatment. A SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other important medical event as per medical or scientific judgment
Time Frame: Up to Week 148
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF-based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Participants
  Any non-SAE (>=2%) | 307 | 304
  Any SAE | 57 | 44

16. Secondary Outcome: Number of Participants With AEs by Their Severity Grades: Up to Week 48
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Adverse events were evaluated by the investigator and graded according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) toxicity scales from Grade 1 to 5 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening, 5=Death). The higher the grade, the more severe the symptoms. Number of participants with adverse events by maximum grade have been presented.
Time Frame: Up to Week 48
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Participants
  Grade 1 | 102 | 94
  Grade 2 | 170 | 177
  Grade 3 | 19 | 15
  Grade 4 | 3 | 6
  Grade 5 | 1 | 0

17. Secondary Outcome: Number of Participants Randomized to TBR Arm Receiving TDF-based Regimen With AEs by Their Severity Grades: Up to Week 48
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Adverse events were evaluated by the investigator and graded according to the DAIDS toxicity scales from Grade 1 to 5 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening, 5=Death). The higher the grade, the more severe the symptoms. Number of TDF-based regimen participants with adverse events by maximum grade have been presented.
Time Frame: Up to Week 48
Population: Safety Population. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen." Data not collected post week 48 as the participant withdrew from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Participants
  Grade 1 | 0
  Grade 2 | 1
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

18. Secondary Outcome: Number of Participants With AEs by Their Severity Grades: Up to Week 144
Description: as for outcome 16
Time Frame: Up to Week 144
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Participants
  Grade 1 | 57 | 65
  Grade 2 | 217 | 208
  Grade 3 | 50 | 54
  Grade 4 | 9 | 8
  Grade 5 | 3 | 0

19. Secondary Outcome: Number of Participants Who Discontinued the Treatment Due to AEs: Up to Week 48
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Number of participants who discontinued the treatment due to adverse events have been presented.
Time Frame: Up to Week 48
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Participants | 13 | 2

20. Secondary Outcome: Number of Participants Randomized to TBR Arm Receiving TDF-based Regimen Who Discontinued the Treatment Due to AEs: Up to Week 48
Description: as for outcome 19
Time Frame: Up to Week 48
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Participants | 0

21. Secondary Outcome: Number of Participants Who Discontinued the Treatment Due to AEs: Up to Week 144
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment.
Time Frame: Up to Week 144
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF-based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Participants | 23 | 7

22. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Hematology Toxicities: Up to Week 48
Description: Blood samples were collected up to Week 48 for the analysis of hematology parameters-platelet count, neutrophils, hemoglobin and leukocytes. Any abnormality in hematology parameters were evaluated according to the DAIDS toxicity scale from Grade 1 to 4: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening). The higher the grade, the more severe the symptoms. Only those participants with maximum post-Baseline emergent hematology toxicities in any of the hematology parameters have been presented.
Time Frame: Up to Week 48
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Participants
  Hemoglobin, Grade 1 | 3 | 0
  Hemoglobin, Grade 2 | 0 | 0
  Hemoglobin, Grade 3 | 0 | 0
  Hemoglobin, Grade 4 | 0 | 0
  Leukocytes, Grade 1 | 1 | 1
  Leukocytes, Grade 2 | 1 | 0
  Leukocytes, Grade 3 | 0 | 0
  Leukocytes, Grade 4 | 0 | 0
  Neutrophils, Grade 1 | 3 | 4
  Neutrophils, Grade 2 | 2 | 4
  Neutrophils, Grade 3 | 0 | 0
  Neutrophils, Grade 4 | 1 | 0
  Platelets, Grade 1 | 6 | 5
  Platelets, Grade 2 | 1 | 1
  Platelets, Grade 3 | 0 | 0
  Platelets, Grade 4 | 0 | 0

23. Secondary Outcome: Number of Participants Randomized to TBR Arm Receiving TDF-based Regimen With Maximum Post-Baseline Emergent Hematology Toxicities: Up to Week 36
Description: Blood samples were collected up to the Week 36 visit for the analysis of hematology parameters-platelet count, neutrophils, hemoglobin and leukocytes. Any abnormality in hematology parameters were evaluated according to the DAIDS toxicity scale from Grade 1 to 4: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening). The higher the grade, the more severe the symptoms. Only those TDF-based regimen participants with maximum post-Baseline emergent hematology toxicities in any of the hematology parameters have been presented.
Time Frame: Up to Week 36
Population: Safety Population. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen." Data not collected post week 36 as the participant withdrew from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Participants
  Hemoglobin, Grade 1 | 0
  Hemoglobin, Grade 2 | 0
  Hemoglobin, Grade 3 | 0
  Hemoglobin, Grade 4 | 0
  Leukocytes, Grade 1 | 0
  Leukocytes, Grade 2 | 0
  Leukocytes, Grade 3 | 0
  Leukocytes, Grade 4 | 0
  Neutrophils, Grade 1 | 0
  Neutrophils, Grade 2 | 0
  Neutrophils, Grade 3 | 0
  Neutrophils, Grade 4 | 0
  Platelets, Grade 1 | 0
  Platelets, Grade 2 | 0
  Platelets, Grade 3 | 0
  Platelets, Grade 4 | 0

24. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Hematology Toxicities: Up to Week 144
Description: Blood samples were collected up to Week 144 for the analysis of hematology parameters-platelet count, neutrophils, hemoglobin and leukocytes. Any abnormality in hematology parameters are were evaluated according to the DAIDS toxicity scale from Grade 1 to 4: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening). The higher the grade, the more severe the symptoms.
Time Frame: Up to Week 144
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Participants
  Hemoglobin, Grade 1 | 7 | 2
  Hemoglobin, Grade 2 | 1 | 2
  Hemoglobin, Grade 3 | 0 | 0
  Hemoglobin, Grade 4 | 0 | 0
  Leukocytes, Grade 1 | 2 | 4
  Leukocytes, Grade 2 | 1 | 0
  Leukocytes, Grade 3 | 1 | 0
  Leukocytes, Grade 4 | 0 | 0
  Neutrophils, Grade 1 | 5 | 5
  Neutrophils, Grade 2 | 3 | 8
  Neutrophils, Grade 3 | 0 | 0
  Neutrophils, Grade 4 | 2 | 2
  Platelets, Grade 1 | 8 | 7
  Platelets, Grade 2 | 2 | 1
  Platelets, Grade 3 | 0 | 0
  Platelets, Grade 4 | 0 | 0

25. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Clinical Chemistry Toxicities: Up to Week 48
Description: Blood samples were collected up to Week 48 for the analysis of clinical chemistry parameters: alanine aminotransferase (ALT), albumin, alkaline phosphate (ALP), aspartate aminotransferase (AST), bilirubin, carbon dioxide (CO2), cholesterol, creatinine kinase (CK), creatinine, direct bilirubin, glomerular filtration rate (GFR) from creatinine adjusted for body surface area (BSA), GFR from cystatin C adjusted using chronic kidney disease-epidemiology collaboration (CKD-EPI), hypercalcemia, hyperglycemia, hyperkalemia, hypernatremia, hypocalcemia, hypoglycemia, hypokalemia, hyponatremia, low density lipoprotein (LDL) cholesterol, phosphate and triglycerides. Any abnormality in clinical chemistry parameters were evaluated according to the DAIDS toxicity scale From Grade 1 to 4: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening). The higher the grade, the more severe the symptoms.
Time Frame: Up to Week 48
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Participants
  ALT, Grade 1 | 24 | 18
  ALT, Grade 2 | 6 | 4
  ALT, Grade 3 | 1 | 1
  ALT, Grade 4 | 0 | 0
  Albumin, Grade 1 | 1 | 0
  Albumin, Grade 2 | 0 | 0
  Albumin, Grade 3 | 0 | 0
  Albumin, Grade 4 | 0 | 0
  ALP, Grade 1 | 2 | 0
  ALP, Grade 2 | 0 | 0
  ALP, Grade 3 | 0 | 0
  ALP, Grade 4 | 0 | 0
  AST, Grade 1 | 21 | 29
  AST, Grade 2 | 7 | 4
  AST, Grade 3 | 1 | 0
  AST, Grade 4 | 1 | 0
  Bilirubin, Grade 1 | 17 | 7
  Bilirubin, Grade 2 | 5 | 2
  Bilirubin, Grade 3 | 1 | 1
  Bilirubin, Grade 4 | 0 | 0
  CO2, Grade 1 | 73 | 70
  CO2, Grade 2 | 1 | 1
  CO2, Grade 3 | 0 | 0
  CO2, Grade 4 | 0 | 0
  Cholesterol, Grade 1 | 27 | 52
  Cholesterol, Grade 2 | 12 | 19
  Cholesterol, Grade 3 | 1 | 0
  Cholesterol, Grade 4 | 0 | 0
  CK, Grade 1 | 28 | 19
  CK, Grade 2 | 4 | 9
  CK, Grade 3 | 9 | 8
  CK, Grade 4 | 6 | 5
  Creatinine, Grade 1 | 16 | 7
  Creatinine, Grade 2 | 3 | 1
  Creatinine, Grade 3 | 0 | 0
  Creatinine, Grade 4 | 0 | 0
  Direct bilirubin, Grade 1 | 0 | 0
  Direct bilirubin, Grade 2 | 0 | 0
  Direct bilirubin, Grade 3 | 8 | 1
  Direct bilirubin, Grade 4 | 0 | 0
  GFR from creatinine adjusted using CKD EPI,Grade 1 | 0 | 0
  GFR from creatinine adjusted using CKD EPI,Grade 2 | 135 | 83
  GFR from creatinine adjusted using CKD EPI,Grade 3 | 26 | 13
  GFR from creatinine adjusted using CKD EPI,Grade 4 | 0 | 0
  GFR from cystatin C adjusted using CKD-EPI,Grade 1 | 0 | 0
  GFR from cystatin C adjusted using CKD-EPI,Grade 2 | 52 | 66
  GFR from cystatin C adjusted using CKD-EPI,Grade 3 | 5 | 4
  GFR from cystatin C adjusted using CKD-EPI,Grade 4 | 1 | 0
  Hypercalcemia, Grade 1 | 7 | 3
  Hypercalcemia, Grade 2 | 0 | 0
  Hypercalcemia, Grade 3 | 0 | 0
  Hypercalcemia, Grade 4 | 0 | 0
  Hyperglycemia, Grade 1 | 56 | 64
  Hyperglycemia, Grade 2 | 21 | 19
  Hyperglycemia, Grade 3 | 2 | 2
  Hyperglycemia, Grade 4 | 0 | 0
  Hyperkalemia, Grade 1 | 0 | 2
  Hyperkalemia, Grade 2 | 2 | 0
  Hyperkalemia, Grade 3 | 0 | 0
  Hyperkalemia, Grade 4 | 0 | 0
  Hypernatremia, Grade 1 | 1 | 1
  Hypernatremia, Grade 2 | 0 | 0
  Hypernatremia, Grade 3 | 0 | 0
  Hypernatremia, Grade 4 | 0 | 0
  Hypocalcemia, Grade 1 | 8 | 1
  Hypocalcemia, Grade 2 | 0 | 1
  Hypocalcemia, Grade 3 | 0 | 0
  Hypocalcemia, Grade 4 | 0 | 0
  Hypoglycemia, Grade 1 | 5 | 6
  Hypoglycemia, Grade 2 | 3 | 2
  Hypoglycemia, Grade 3 | 0 | 0
  Hypoglycemia, Grade 4 | 0 | 0
  Hypokalemia, Grade 1 | 7 | 1
  Hypokalemia, Grade 2 | 1 | 0
  Hypokalemia, Grade 3 | 0 | 0
  Hypokalemia, Grade 4 | 0 | 0
  Hyponatremia, Grade 1 | 8 | 13
  Hyponatremia, Grade 2 | 0 | 2
  Hyponatremia, Grade 3 | 0 | 0
  Hyponatremia, Grade 4 | 0 | 0
  LDL cholesterol, Grade 1 | 28 | 35
  LDL cholesterol, Grade 2 | 13 | 15
  LDL cholesterol, Grade 3 | 6 | 3
  LDL cholesterol, Grade 4 | 0 | 0
  Phosphate, Grade 1 | 38 | 47
  Phosphate, Grade 2 | 2 | 7
  Phosphate, Grade 3 | 0 | 0
  Phosphate, Grade 4 | 0 | 0
  Triglycerides, Grade 1 | 34 | 48
  Triglycerides, Grade 2 | 4 | 11
  Triglycerides, Grade 3 | 4 | 4
  Triglycerides, Grade 4 | 4 | 0

26. Secondary Outcome: Number of Participants Randomized to TBR Arm Receiving TDF-based Regimen With Maximum Post-Baseline Emergent Clinical Chemistry Toxicities: Up to Week 36
Description: samples were collected up to the Week 36 visit for the analysis of clinical chemistry parameters: alanine aminotransferase (ALT), albumin, alkaline phosphate (ALP), aspartate aminotransferase (AST), bilirubin, carbon dioxide (CO2), cholesterol, creatinine kinase (CK), creatinine, direct bilirubin, glomerular filtration rate (GFR) from creatinine adjusted using chronic kidney disease-epidemiology collaboration (CKD-EPI), GFR from cystatin C adjusted using CKD-EPI, hypercalcemia, hyperglycemia, hyperkalemia, hypernatremia, hypocalcemia, hypoglycemia, hypokalemia, hyponatremia, low density lipoprotein (LDL) cholesterol, phosphate and triglycerides. Any abnormality in clinical chemistry parameters were evaluated according to the DAIDS toxicity scale From Grade 1 to 4: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening). The higher the grade, the more severe the symptoms.
Time Frame: Up to Week 36
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Participants
  ALT, Grade 1 | 0
  ALT, Grade 2 | 0
  ALT, Grade 3 | 0
  ALT, Grade 4 | 0
  Albumin, Grade 1 | 0
  Albumin, Grade 2 | 0
  Albumin, Grade 3 | 0
  Albumin, Grade 4 | 0
  ALP, Grade 1 | 0
  ALP, Grade 2 | 0
  ALP, Grade 3 | 0
  ALP, Grade 4 | 0
  AST, Grade 1 | 0
  AST, Grade 2 | 0
  AST, Grade 3 | 0
  AST, Grade 4 | 0
  Bilirubin, Grade 1 | 0
  Bilirubin, Grade 2 | 0
  Bilirubin, Grade 3 | 0
  Bilirubin, Grade 4 | 0
  CO2, Grade 1 | 0
  CO2, Grade 2 | 0
  CO2, Grade 3 | 0
  CO2, Grade 4 | 0
  Cholesterol, Grade 1 | 0
  Cholesterol, Grade 2 | 0
  Cholesterol, Grade 3 | 0
  Cholesterol, Grade 4 | 0
  CK, Grade 1 | 0
  CK, Grade 2 | 0
  CK, Grade 3 | 0
  CK, Grade 4 | 0
  Creatinine, Grade 1 | 0
  Creatinine, Grade 2 | 0
  Creatinine, Grade 3 | 0
  Creatinine, Grade 4 | 0
  Direct bilirubin, Grade 1 | 0
  Direct bilirubin, Grade 2 | 0
  Direct bilirubin, Grade 3 | 0
  Direct bilirubin, Grade 4 | 0
  GFR from creatinine adjusted using CKD EPI,Grade 1 | 0
  GFR from creatinine adjusted using CKD EPI,Grade 2 | 0
  GFR from creatinine adjusted using CKD EPI,Grade 3 | 0
  GFR from creatinine adjusted using CKD EPI,Grade 4 | 0
  GFR from cystatin C adjusted using CKD-EPI,Grade 1 | 0
  GFR from cystatin C adjusted using CKD-EPI,Grade 2 | 0
  GFR from cystatin C adjusted using CKD-EPI,Grade 3 | 0
  GFR from cystatin C adjusted using CKD-EPI,Grade 4 | 0
  Hypercalcemia, Grade 1 | 0
  Hypercalcemia, Grade 2 | 0
  Hypercalcemia, Grade 3 | 0
  Hypercalcemia, Grade 4 | 0
  Hyperglycemia, Grade 1 | 0
  Hyperglycemia, Grade 2 | 0
  Hyperglycemia, Grade 3 | 0
  Hyperglycemia, Grade 4 | 0
  Hyperkalemia, Grade 1 | 0
  Hyperkalemia, Grade 2 | 0
  Hyperkalemia, Grade 3 | 0
  Hyperkalemia, Grade 4 | 0
  Hypernatremia, Grade 1 | 0
  Hypernatremia, Grade 2 | 0
  Hypernatremia, Grade 3 | 0
  Hypernatremia, Grade 4 | 0
  Hypocalcemia, Grade 1 | 0
  Hypocalcemia, Grade 2 | 0
  Hypocalcemia, Grade 3 | 0
  Hypocalcemia, Grade 4 | 0
  Hypoglycemia, Grade 1 | 0
  Hypoglycemia, Grade 2 | 0
  Hypoglycemia, Grade 3 | 0
  Hypoglycemia, Grade 4 | 0
  Hypokalemia, Grade 1 | 0
  Hypokalemia, Grade 2 | 0
  Hypokalemia, Grade 3 | 0
  Hypokalemia, Grade 4 | 0
  Hyponatremia, Grade 1 | 0
  Hyponatremia, Grade 2 | 0
  Hyponatremia, Grade 3 | 0
  Hyponatremia, Grade 4 | 0
  LDL cholesterol, Grade 1 | 0
  LDL cholesterol, Grade 2 | 0
  LDL cholesterol, Grade 3 | 0
  LDL cholesterol, Grade 4 | 0
  Phosphate, Grade 1 | 0
  Phosphate, Grade 2 | 0
  Phosphate, Grade 3 | 0
  Phosphate, Grade 4 | 0
  Triglycerides, Grade 1 | 1
  Triglycerides, Grade 2 | 0
  Triglycerides, Grade 3 | 0
  Triglycerides, Grade 4 | 0

27. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Clinical Chemistry Toxicities: Up to Week 144
Description: Blood samples were collected up to Week 144 for the analysis of clinical chemistry parameters: ALT, albumin, ALP, AST, bilirubin, CO2, cholesterol, CK, creatinine, direct bilirubin, GFR from creatinine adjusted for BSA, GFR from cystatin C adjusted using CKD-EPI, hypercalcemia, hyperglycemia, hyperkalemia, hypernatremia, hypocalcemia, hypoglycemia, hypokalemia, hyponatremia, LDL cholesterol, phosphate triglycerides and lactate dehydrogenase. Any abnormality in clinical chemistry parameters were evaluated according to the DAIDS toxicity scale From Grade 1 to 4: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening). The higher the grade, the more severe the symptoms.
Time Frame: Up to Week 144
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Participants
  ALT, Grade 1 | 55 | 49
  ALT, Grade 2 | 11 | 9
  ALT, Grade 3 | 5 | 3
  ALT, Grade 4 | 0 | 1
  Albumin, Grade 1 | 1 | 0
  Albumin, Grade 2 | 2 | 0
  Albumin, Grade 3 | 0 | 0
  Albumin, Grade 4 | 0 | 0
  ALP, Grade 1 | 6 | 0
  ALP, Grade 2 | 0 | 0
  ALP, Grade 3 | 0 | 1
  ALP, Grade 4 | 0 | 0
  AST, Grade 1 | 34 | 45
  AST, Grade 2 | 13 | 9
  AST, Grade 3 | 3 | 0
  AST, Grade 4 | 3 | 3
  Bilirubin, Grade 1 | 24 | 12
  Bilirubin, Grade 2 | 9 | 4
  Bilirubin, Grade 3 | 3 | 1
  Bilirubin, Grade 4 | 0 | 0
  CO2, Grade 1 | 110 | 97
  CO2, Grade 2 | 2 | 4
  CO2, Grade 3 | 1 | 0
  CO2, Grade 4 | 0 | 0
  Cholesterol, Grade 1 | 42 | 70
  Cholesterol, Grade 2 | 26 | 34
  Cholesterol, Grade 3 | 1 | 2
  Cholesterol, Grade 4 | 0 | 0
  CK, Grade 1 | 41 | 30
  CK, Grade 2 | 12 | 13
  CK, Grade 3 | 12 | 12
  CK, Grade 4 | 10 | 10
  Creatinine, Grade 1 | 21 | 12
  Creatinine, Grade 2 | 5 | 2
  Creatinine, Grade 3 | 1 | 1
  Creatinine, Grade 4 | 0 | 0
  Direct bilirubin, Grade 1 | 0 | 0
  Direct bilirubin, Grade 2 | 0 | 0
  Direct bilirubin, Grade 3 | 13 | 3
  Direct bilirubin, Grade 4 | 0 | 0
  GFR from creatinine adjusted using CKD EPI,Grade 1 | 0 | 0
  GFR from creatinine adjusted using CKD EPI,Grade 2 | 165 | 101
  GFR from creatinine adjusted using CKD EPI,Grade 3 | 38 | 24
  GFR from creatinine adjusted using CKD EPI,Grade 4 | 0 | 1
  GFR from cystatin C adjusted using CKD-EPI,Grade 1 | 0 | 0
  GFR from cystatin C adjusted using CKD-EPI,Grade 2 | 169 | 183
  GFR from cystatin C adjusted using CKD-EPI,Grade 3 | 46 | 58
  GFR from cystatin C adjusted using CKD-EPI,Grade 4 | 1 | 1
  Hypercalcemia, Grade 1 | 8 | 9
  Hypercalcemia, Grade 2 | 0 | 0
  Hypercalcemia, Grade 3 | 0 | 0
  Hypercalcemia, Grade 4 | 0 | 0
  Hyperglycemia, Grade 1 | 73 | 77
  Hyperglycemia, Grade 2 | 40 | 31
  Hyperglycemia, Grade 3 | 4 | 4
  Hyperglycemia, Grade 4 | 0 | 0
  Hyperkalemia, Grade 1 | 3 | 2
  Hyperkalemia, Grade 2 | 2 | 1
  Hyperkalemia, Grade 3 | 0 | 0
  Hyperkalemia, Grade 4 | 0 | 0
  Hypernatremia, Grade 1 | 4 | 3
  Hypernatremia, Grade 2 | 1 | 0
  Hypernatremia, Grade 3 | 0 | 0
  Hypernatremia, Grade 4 | 0 | 0
  Hypocalcemia, Grade 1 | 14 | 5
  Hypocalcemia, Grade 2 | 1 | 2
  Hypocalcemia, Grade 3 | 0 | 0
  Hypocalcemia, Grade 4 | 0 | 0
  Hypoglycemia, Grade 1 | 9 | 10
  Hypoglycemia, Grade 2 | 4 | 3
  Hypoglycemia, Grade 3 | 0 | 0
  Hypoglycemia, Grade 4 | 0 | 0
  Hypokalemia, Grade 1 | 10 | 7
  Hypokalemia, Grade 2 | 3 | 0
  Hypokalemia, Grade 3 | 1 | 0
  Hypokalemia, Grade 4 | 0 | 0
  Hyponatremia, Grade 1 | 21 | 26
  Hyponatremia, Grade 2 | 0 | 2
  Hyponatremia, Grade 3 | 0 | 0
  Hyponatremia, Grade 4 | 0 | 0
  LDL cholesterol, Grade 1 | 41 | 56
  LDL cholesterol, Grade 2 | 19 | 24
  LDL cholesterol, Grade 3 | 8 | 9
  LDL cholesterol, Grade 4 | 0 | 0
  Phosphate, Grade 1 | 61 | 71
  Phosphate, Grade 2 | 3 | 9
  Phosphate, Grade 3 | 0 | 0
  Phosphate, Grade 4 | 0 | 0
  Triglycerides, Grade 1 | 60 | 77
  Triglycerides, Grade 2 | 6 | 15
  Triglycerides, Grade 3 | 6 | 5
  Triglycerides, Grade 4 | 4 | 2
  Lactate Dehydrogenase Grade 1 | 0 | 1
  Lactate Dehydrogenase Grade 2 | 0 | 0
  Lactate Dehydrogenase Grade 3 | 0 | 0
  Lactate Dehydrogenase Grade 4 | 0 | 0

28. Secondary Outcome: Change From Baseline in Renal Biomarkers- Urine Albumin/Creatinine (UA/C) Ratio and Urine Protein/Creatinine (UP/C) Ratio at Weeks 24 and 48
Description: Urine samples were collected at Baseline, Week 24 and Week 48. Baseline is defined as Day 1. Change from Baseline in UA/C was calculated as UA/C ratio at post-Baseline visit minus UA/C ratio calculated at Baseline. Estimated geometric mean adjusted ratio (each visit over Baseline) and 95% CI have been presented. Change from Baseline in UP/C and UA/C was calculated as UP/C and UA/C ratio at post-Baseline visit minus UP/C and UA/C ratio calculated at Baseline, respectively. Estimated geometric mean adjusted ratio (each visit over Baseline) and 95% CI have been presented. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at weeks 24 and 48
Population: Safety Population. Total of 741 participants were analyzed but 740 participants are presented in this Outcome Measure and 1 participant is presented separately in next Outcome Measure. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Ratio
  UA/C, Week 24, n=235, 230: number analyzed (Participants) | 235 | 230
  UA/C, Week 24, n=235, 230 | 1.080 [1.007 to 1.158] | 1.022 [0.956 to 1.091]
  UA/C, Week 48, n=230, 224: number analyzed (Participants) | 230 | 224
  UA/C, Week 48, n=230, 224 | 1.125 [1.036 to 1.222] | 1.059 [0.963 to 1.165]
  UP/C, Week 24, n=267, 261: number analyzed (Participants) | 267 | 261
  UP/C, Week 24, n=267, 261 | 0.955 [0.917 to 0.995] | 0.976 [0.937 to 1.016]
  UP/C, Week 48, n=261, 257: number analyzed (Participants) | 261 | 257
  UP/C, Week 48, n=261, 257 | 0.971 [0.926 to 1.018] | 1.016 [0.964 to 1.070]
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.257, Mixed Model Repeated Measures; Treatment ratio = 1.057, 95% CI 2-sided [0.960 to 1.164] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for UA/C at Week 24 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.350, Mixed Model Repeated Measures; Treatment ratio = 1.062, 95% CI 2-sided [0.936 to 1.205] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for UA/C at Week 48 has been presented
Statistical Analysis 3: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.473, Mixed Model Repeated Measures; Treatment ratio = 0.979, 95% CI 2-sided [0.924 to 1.037] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for UP/C at Week 24 has been presented
Statistical Analysis 4: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.212, Mixed Model Repeated Measures; Treatment ratio = 0.956, 95% CI 2-sided [0.891 to 1.026] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for UP/C at Week 48 has been presented

29. Secondary Outcome: Change From Baseline in Renal Biomarkers- UA/C Ratio and UP/C Ratio at Weeks 24 and 48 in Participants Randomized to TBR Receiving TDF-based Regimen
Description: Urine samples were collected at Baseline, Week 24 and Week 48 to assess renal biomarkers - urine albumin/creatinine ratio and urine protein/creatinine ratio. Baseline was defined as the latest pre-dose assessment value with a non-missing value. (Day 1). Change from Baseline in UA/C was calculated as UA/C ratio at post-Baseline visit minus UA/C ratio calculated at Baseline. Change from Baseline in UP/C was calculated as UP/C ratio at post-Baseline visit minus UP/C ratio calculated at Baseline. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at weeks 24 and 48
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Data not collected post week 48 as the participant withdrew from the study.
Measure: Number; unit: Ratio
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Ratio
  UA/C, Week 24, n=1 | 0
  UA/C, Week 48, n=0: number analyzed (Participants) | 0
  UP/C, Week 24, n=1 | 0.3
  UP/C, Week 48, n=0: number analyzed (Participants) | 0

30. Secondary Outcome: Change From Baseline in Renal Biomarkers- UA/C Ratio and UP/C Ratio at Weeks 96 and 144
Description: Urine samples were collected at Baseline, Weeks 96 and 144. Baseline is defined as Day 1. Change from Baseline in UA/C is defined as UA/C ratio at post-Baseline visit minus UA/C ratio at Baseline. Change from Baseline in UP/C and UA/C is defined as UP/C and UA/C ratio at post-Baseline visit minus UP/C and UA/C ratio at Baseline, respectively. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen.
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DTG+3TC FDC (Early Switch) | TAF-based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Ratio
  UA/C, Week 96, n=208, 175: number analyzed (Participants) | 208 | 175
  UA/C, Week 96, n=208, 175 | 1.058 [0.974 to 1.149] | 1.075 [0.968 to 1.195]
  UA/C, Week 144, n=202, 179: number analyzed (Participants) | 202 | 179
  UA/C, Week 144, n=202, 179 | 1.203 [1.093 to 1.324] | 1.200 [1.051 to 1.371]
  UP/C, Week 96, n=245, 206: number analyzed (Participants) | 245 | 206
  UP/C, Week 96, n=245, 206 | 1.048 [0.997 to 1.102] | 1.105 [1.044 to 1.169]
  UP/C, Week 144, n=237, 220: number analyzed (Participants) | 237 | 220
  UP/C, Week 144, n=237, 220 | 1.182 [1.121 to 1.247] | 1.188 [1.104 to 1.278]
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.700, Mixed Model Repeated Measures; Treatment ratio = 0.977, 95% CI 2-sided [0.866 to 1.102] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for UA/C at Week 96 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.700, Mixed Model Repeated Measures; Treatment ratio = 0.971, 95% CI 2-sided [0.835 to 1.129] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for UA/C at Week 144 has been presented
Statistical Analysis 3: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.356, Mixed Model Repeated Measures; Treatment ratio = 0.969, 95% CI 2-sided [0.907 to 1.036] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for UP/C at Week 96 has been presented
Statistical Analysis 4: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.814, Mixed Model Repeated Measures; Treatment ratio = 0.991, 95% CI 2-sided [0.916 to 1.071] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for UP/C at Week 144 has been presented

31. Secondary Outcome: Change From Baseline in Renal Biomarkers- Urine Beta-2 Microglobulin/Urine Creatinine Ratio at Weeks 24 and 48
Description: Urine biomarker samples were collected at Baseline, Weeks 24 and 48 to assess urine beta-2 microglobulin/urine creatinine. Geometric mean ratio (visit divided by Baseline) and 95% CI of geometric mean ratio has been presented. Baseline (Day 1) value was the value from the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline in urine beta-2-microglobulin/urine creatinine was calculated as urine beta-2-microglobulin/urine creatinine ratio at post-Baseline visit minus urine beta-2-microglobulin/urine creatinine ratio calculated at Baseline. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at weeks 24 and 48
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Ratio
  Week 24, n=136, 141: number analyzed (Participants) | 136 | 141
  Week 24, n=136, 141 | 0.991 [0.899 to 1.093] | 1.034 [0.931 to 1.149]
  Week 48, n=126, 141: number analyzed (Participants) | 126 | 141
  Week 48, n=126, 141 | 0.973 [0.870 to 1.088] | 0.922 [0.832 to 1.022]
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.560, Mixed Model Repeated Measures; Treatment ratio = 0.958, 95% CI 2-sided [0.830 to 1.106] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for Urine beta-2 microglobulin/urine creatinine at Week 24 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.489, Mixed Model Repeated Measures; Treatment ratio = 1.055, 95% CI 2-sided [0.906 to 1.229] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for Urine beta-2 microglobulin/urine creatinine at Week 48 has been presented

32. Secondary Outcome: Change From Baseline in Renal Biomarkers- Urine Beta-2 Microglobulin/Urine Creatinine Ratio at Weeks 24 and 48 in Participants Randomized to TBR Arm Receiving TDF-based Regimen
Description: Urine biomarker samples were collected to assess urine beta-2 microglobulin/urine creatinine. Baseline (Day 1) value was the value from the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline in urine beta-2-microglobulin/urine creatinine was calculated as urine beta-2-microglobulin/urine creatinine ratio at post-Baseline visit minus urine beta-2-microglobulin/urine creatinine ratio calculated at Baseline. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at weeks 24 and 48
Population: Safety Population. Data was not collected for this arm. Data not collected post week 48 as the participant withdrew from the study.
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 0

33. Secondary Outcome: Change From Baseline in Renal Biomarkers- Urine Beta-2 Microglobulin/Urine Creatinine Ratio at Weeks 96 and 144
Description: Urine biomarker samples were collected at Baseline, Weeks 96 and 144 to assess urine beta-2 microglobulin/urine creatinine. Baseline (Day 1) value is the value from the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline in urine beta-2-microglobulin/urine creatinine is defined as urine beta-2-microglobulin/urine creatinine ratio at post-Baseline visit minus urine beta-2-microglobulin/urine creatinine ratio at Baseline. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen.
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: Safety Population. Total of 741 participants were analyzed but 740 participants are presented in this Outcome Measure and 1 participant is presented separately in next Outcome Measure. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category title)
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DTG+3TC FDC (Early Switch) | TAF-based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Ratio
  Week 96, n=109, 107: number analyzed (Participants) | 109 | 107
  Week 96, n=109, 107 | 1.080 [0.931 to 1.253] | 0.986 [0.844 to 1.152]
  Week 144, n=101, 97: number analyzed (Participants) | 101 | 97
  Week 144, n=101, 97 | 0.904 [0.768 to 1.065] | 0.958 [0.808 to 1.136]
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.081, Mixed Model Repeated Measures; Treatment ratio = 1.165, 95% CI 2-sided [0.981 to 1.384] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for Urine beta-2 microglobulin/urine creatinine at Week 96 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.834, Mixed Model Repeated Measures; Treatment ratio = 0.981, 95% CI 2-sided [0.819 to 1.175] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for Urine beta-2 microglobulin/urine creatinine at Week 144 has been presented

34. Secondary Outcome: Change From Baseline in Renal Biomarkers- Urine Phosphate at Weeks 24 and 48
Description: Urine biomarker samples were collected at Baseline and at Weeks 24 and 48 to assess urine phosphate. Geometric mean ratio (visit divided by Baseline) and 95% CI of geometric mean ratio has been presented. Baseline (Day 1) value was the value from the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline in urine phosphate was calculated as urine phosphate at post-Baseline visit minus urine phosphate calculated at Baseline. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at weeks 24 and 48
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Ratio
  Week 24, n=348, 352: number analyzed (Participants) | 348 | 352
  Week 24, n=348, 352 | 0.955 [0.888 to 1.028] | 0.940 [0.871 to 1.014]
  Week 48, n=342, 340: number analyzed (Participants) | 342 | 340
  Week 48, n=342, 340 | 0.969 [0.892 to 1.052] | 0.970 [0.900 to 1.044]
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.758, Mixed Model Repeated Measures; Treatment ratio = 1.017, 95% CI 2-sided [0.915 to 1.130] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for Urine phosphate at Week 24 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.985, Mixed Model Repeated Measures; Treatment ratio = 0.999, 95% CI 2-sided [0.894 to 1.116] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for Urine phosphate at Week 48 has been presented

35. Secondary Outcome: Change From Baseline in Renal Biomarkers- Urine Phosphate at Weeks 24 and 48 in Participants Randomized to TBR Arm Receiving TDF-based Regimen
Description: Urine biomarker samples were collected to assess urine phosphate. Baseline (Day 1) value was the value from the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline in urine phosphate was calculated as urine phosphate at post-Baseline visit minus urine phosphate calculated at Baseline. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at weeks 24 and 48
Population: as for outcome 29
Measure: Number; unit: Ratio
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Ratio
  Week 24, n=1 | 2.9
  Week 48, n=0: number analyzed (Participants) | 0

36. Secondary Outcome: Change From Baseline in Renal Biomarkers- Urine Phosphate at Weeks 96 and 144
Description: Urine biomarker samples were collected at Baseline, Weeks 96 and 144 to assess urine phosphate. Baseline (Day 1) value is the value from the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline in urine phosphate is defined as urine phosphate at post-Baseline visit minus urine phosphate at Baseline. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Ratio
  Week 96, n=312, 286: number analyzed (Participants) | 312 | 286
  Week 96, n=312, 286 | 0.960 [0.871 to 1.057] | 0.978 [0.882 to 1.085]
  Week 144, n=313, 298: number analyzed (Participants) | 313 | 298
  Week 144, n=313, 298 | 0.890 [0.805 to 0.985] | 0.912 [0.825 to 1.007]
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.806, Mixed Model Repeated Measures; Treatment ratio = 1.015, 95% CI 2-sided [0.904 to 1.139] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for Urine phosphate at Week 96 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.745, Mixed Model Repeated Measures; Treatment ratio = 1.019, 95% CI 2-sided [0.909 to 1.142] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for Urine phosphate at Week 144 has been presented

37. Secondary Outcome: Change From Baseline in Renal Biomarkers- Urine Retinol Binding Protein 4/Urine Creatinine at Weeks 24 and 48
Description: Urine biomarker samples were collected at Baseline, Weeks 24 and 48 to assess urine retinol binding protein 4/urine creatinine. Geometric mean ratio (visit divided by Baseline) and 95% CI of geometric mean ratio has been presented. Baseline (Day 1) value was the value from the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline in Urine retinol binding protein 4/urine creatinine ratio was calculated as Urine retinol binding protein 4/urine creatinine ratio at post-Baseline visit minus Urine retinol binding protein 4/urine creatinine ratio calculated at Baseline. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at weeks 24 and 48
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Ratio
  Week 24, n=344, 343: number analyzed (Participants) | 344 | 343
  Week 24, n=344, 343 | 0.860 [0.790 to 0.936] | 0.920 [0.847 to 0.999]
  Week 48, n=340, 335: number analyzed (Participants) | 340 | 335
  Week 48, n=340, 335 | 1.063 [0.992 to 1.139] | 1.068 [0.996 to 1.144]
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.264, Mixed Model Reported Measures; Treatment ratio = 0.935, 95% CI 2-sided [0.830 to 1.052] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for Urine retinol binding protein 4/urine creatinine at Week 24 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.932, Mixed Model Repeated Measures; Treatment ratio = 0.996, 95% CI 2-sided [0.903 to 1.098] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for Urine retinol binding protein 4/urine creatinine at Week 48 has been presented

38. Secondary Outcome: Change From Baseline in Renal Biomarkers- Urine Retinol Binding Protein 4/Urine Creatinine at Weeks 24 and 48 in Participants Randomized to TBR Arm Receiving TDF-based Regimen
Description: Urine biomarker samples were collected to assess urine retinol binding protein 4/urine creatinine. Baseline (Day 1) value was the value from the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline in urine retinol binding protein 4/urine creatinine was calculated as urine retinol binding protein 4/urine creatinine ratio at post-Baseline visit minus urine retinol binding protein 4/urine creatinine ratio calculated at Baseline. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at weeks 24 and 48
Population: as for outcome 29
Measure: Number; unit: Ratio
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Ratio
  Week 24, n=1 | 1.04
  Week 48, n=0: number analyzed (Participants) | 0

39. Secondary Outcome: Change From Baseline in Renal Biomarkers- Urine Retinol Binding Protein 4/Urine Creatinine at Weeks 96 and 144
Description: Urine biomarker samples were collected at Baseline, Weeks 96 and 144 to assess urine retinol binding protein 4/urine creatinine. Baseline (Day 1) value is the value from the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline in Urine retinol binding protein 4/urine creatinine ratio is defined as Urine retinol binding protein 4/urine creatinine ratio at post-Baseline visit minus Urine retinol binding protein 4/urine creatinine ratio at Baseline. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- DTG+3TC FDC (Early Switch): Participants who were on a stable TBR and who had an HIV-1 ribonucleic acid (RNA) <50 copies per millilter (c/mL) at the time of screening, received fixed dose combination of DTG 50 milligrams (mg) + 3TC 300 mg once daily up to 48 weeks.
- TAF Based Regimen (Early Switch): Participants who were on a stable TBR and who had an HIV-1 RNA<50 c/mL at the time of screening, were continued to receive TBR up to 48 weeks. One participant randomized to the this arm received TDF rather than TAF-and was presented within the "TAF-based regimen" arm for efficacy because the efficacy of TAF and TDF are comparable. However the participant was presented separately under "TDF-based regimen" for Safety because the safety profiles of TDF and TAF differ.
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Ratio
  Week 96, n=310, 282: number analyzed (Participants) | 310 | 282
  Week 96, n=310, 282 | 0.926 [0.845 to 1.014] | 0.851 [0.775 to 0.933]
  Week 144, n=304, 288: number analyzed (Participants) | 304 | 288
  Week 144, n=304, 288 | 1.188 [1.086 to 1.298] | 1.227 [1.109 to 1.359]
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.011, Mixed Model Repeated Measures; Treatment ratio = 1.150, 95% CI 2-sided [1.032 to 1.281] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for Urine retinol binding protein 4/urine creatinine at Week 96 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.895, Mixed Model Repeated Measures; Treatment ratio = 1.007, 95% CI 2-sided [0.905 to 1.121] — Treatment ratio (DTG+3TC/ TAF based regimen) and 95% CI for Urine retinol binding protein 4/urine creatinine at Week 144 has been presented

40. Secondary Outcome: Change From Baseline in Fasting Lipids at Weeks 24 and 48
Description: Blood samples were collected at Baseline (Day 1), Week 24 and Week 48 to assess fasting lipids which included plasma cholesterol, plasma LDL cholesterol, plasma high density lipoprotein (HDL) cholesterol and plasma triglycerides. Baseline value was the value from the latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at weeks 24 and 48
Population: as for outcome 28
Measure: Median (Inter-Quartile Range); unit: Millimoles per liter
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Millimoles per liter
  Plasma cholesterol, Week 24, n=282, 264: number analyzed (Participants) | 282 | 264
  Plasma cholesterol, Week 24, n=282, 264 | -0.325 [-0.750 to 0.150] | 0.000 [-0.400 to 0.400]
  Plasma cholesterol, Week 48, n=275, 263: number analyzed (Participants) | 275 | 263
  Plasma cholesterol, Week 48, n=275, 263 | -0.200 [-0.750 to 0.150] | 0.100 [-0.350 to 0.500]
  Plasma LDL Cholesterol, Week 24, n=282, 264: number analyzed (Participants) | 282 | 264
  Plasma LDL Cholesterol, Week 24, n=282, 264 | -0.210 [-0.570 to 0.130] | -0.060 [-0.340 to 0.410]
  Plasma LDL Cholesterol, Week 48, n=275, 263: number analyzed (Participants) | 275 | 263
  Plasma LDL Cholesterol, Week 48, n=275, 263 | -0.170 [-0.560 to 0.210] | 0.070 [-0.320 to 0.430]
  Plasma Triglycerides, Week 24, n=282, 264: number analyzed (Participants) | 282 | 264
  Plasma Triglycerides, Week 24, n=282, 264 | -0.100 [-0.460 to 0.160] | 0.060 [-0.200 to 0.350]
  Plasma Triglycerides, Week 48, n=275, 263: number analyzed (Participants) | 275 | 263
  Plasma Triglycerides, Week 48, n=275, 263 | -0.100 [-0.440 to 0.160] | 0.100 [-0.280 to 0.380]
  Plasma HDL Cholesterol, Week 24, n=282, 264: number analyzed (Participants) | 282 | 264
  Plasma HDL Cholesterol, Week 24, n=282, 264 | -0.050 [-0.150 to 0.100] | 0.050 [-0.150 to 0.150]
  Plasma HDL Cholesterol, Week 48, n=275, 263: number analyzed (Participants) | 275 | 263
  Plasma HDL Cholesterol, Week 48, n=275, 263 | 0.000 [-0.200 to 0.150] | 0.050 [-0.150 to 0.150]

41. Secondary Outcome: Change From Baseline in Fasting Lipids at Weeks 24 and 48 in Participants Randomized to TBR Arm Receiving TDF-based Regimen
Description: Blood samples were collected at Baseline (Day 1), weeks 24 and 48 visit (participant withdrew from the study at Week 36) to assess fasting lipids which included plasma cholesterol, plasma LDL cholesterol, plasma HDL cholesterol and plasma triglycerides. Baseline value was the value from the latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. Change from Baseline values for fasting lipids in TDF-based regimen participants has been presented. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at weeks 24 and 48
Population: as for outcome 29
Measure: Number; unit: Millimoles per liter
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Millimoles per liter
  Plasma cholesterol, Week 24, n=1 | 0
  Plasma cholesterol, Week 48, n=0: number analyzed (Participants) | 0
  Plasma LDL Cholesterol, Week 24, n=1 | -0.67
  Plasma LDL Cholesterol, Week 48, n=0: number analyzed (Participants) | 0
  Plasma Triglycerides, Week 24, n=1 | 1.36
  Plasma Triglycerides, Week 48, n=0: number analyzed (Participants) | 0
  Plasma HDL Cholesterol, Week 24, n=1 | 0.05
  Plasma HDL Cholesterol, Week 48, n=0: number analyzed (Participants) | 0

42. Secondary Outcome: Change From Baseline in Fasting Lipids at Weeks 96 and 144
Description: Blood samples were collected at Baseline (Day 1), Weeks 96 and 144 to assess fasting lipids which includes plasma cholesterol, plasma LDL cholesterol, plasma HDL cholesterol and plasma triglycerides. Baseline value is the value from the latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen.
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: as for outcome 28
Measure: Median (Inter-Quartile Range); unit: Millimoles per liter
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Millimoles per liter
  Plasma cholesterol, Week 96, n=238, 213: number analyzed (Participants) | 238 | 213
  Plasma cholesterol, Week 96, n=238, 213 | -3.7 [-12.4 to 5.6] | 1.2 [-6.0 to 10.6]
  Plasma cholesterol, Week 144, n=243, 230: number analyzed (Participants) | 243 | 230
  Plasma cholesterol, Week 144, n=243, 230 | -4.0 [-13.0 to 6.4] | 3.8 [-5.0 to 14.5]
  Plasma LDL Cholesterol, Week 96, n=238, 213: number analyzed (Participants) | 238 | 213
  Plasma LDL Cholesterol, Week 96, n=238, 213 | -5.6 [-17.3 to 10.8] | 1.7 [-8.9 to 15.8]
  Plasma LDL Cholesterol, Week 144, n=243, 230: number analyzed (Participants) | 243 | 230
  Plasma LDL Cholesterol, Week 144, n=243, 230 | -5.0 [-16.2 to 10.7] | 4.2 [-9.0 to 20.9]
  Plasma Triglycerides, Week 96, n=238, 213: number analyzed (Participants) | 238 | 213
  Plasma Triglycerides, Week 96, n=238, 213 | -2.1 [-25.8 to 22.2] | 4.9 [-20.0 to 38.9]
  Plasma Triglycerides, Week 144, n=243, 230: number analyzed (Participants) | 243 | 230
  Plasma Triglycerides, Week 144, n=243, 230 | -9.4 [-32.8 to 21.2] | 2.2 [-23.0 to 30.3]
  Plasma HDL Cholesterol, Week 96, n=238, 213: number analyzed (Participants) | 238 | 213
  Plasma HDL Cholesterol, Week 96, n=238, 213 | -3.8 [-13.8 to 8.5] | 0.0 [-10.8 to 13.0]
  Plasma HDL Cholesterol, Week 144, n=243, 230: number analyzed (Participants) | 243 | 230
  Plasma HDL Cholesterol, Week 144, n=243, 230 | -3.8 [-14.3 to 12.0] | 3.8 [-8.0 to 17.4]

43. Secondary Outcome: Number of Participants With Genotypic Resistance: Up to Week 48
Description: Plasma samples were collected for drug resistance testing. Number of participants, who met confirmed virologic withdrawal (CVW) criteria (one plasma HIV-1 RNA >=200 c/mL after Day 1 with immediate prior HIV RNA >=50 c/mL), with genotypic resistance to INSTI, nucleoside reverse transcriptase inhibitor (NRTI), NNRTI and PI was summarized.
Time Frame: Up to Week 48
Population: CVW Population comprised of all participants in the ITT-E Population who had met the derived CVW criteria. One participant randomized to TBR but received TDF-based regimen and was presented within the "TBR (TAF-based regimen) arm" as efficacy of TAF and TDF are comparable.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 0 | 1
Participants
  INSTI |  | 0
  NRTI |  | 0
  NNRTI |  | 0
  PI |  | 0

44. Secondary Outcome: Number of Participants With Genotypic Resistance: Up to Week 144
Description: Plasma samples were collected for drug resistance testing. Number of participants, who meet CVW criteria (one plasma HIV-1 RNA >=200 c/mL after Day 1 with immediate prior HIV RNA >=50 c/mL), with genotypic resistance to INSTI, NRTI, NNRTI and PI are summarized.
Time Frame: Up to Week 144
Population: CVW Population comprises all participants in the ITT-E Population who had met the derived CVW criteria and who had resistance data. One participant randomized to TBR but received TDF-based regimen and was presented within the "TBR (TAF-based regimen) arm" as efficacy of TAF and TDF are comparable.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 0 | 2
Participants
  INSTI |  | 0
  NRTI |  | 0
  NNRTI |  | 0
  PI |  | 0

45. Secondary Outcome: Number of Participants With Phenotypic Resistance: Up to Week 48
Description: Number of participants, who meet CVW criteria (one plasma HIV-1 RNA >=200 c/mL after Day 1 with immediate prior HIV RNA >=50 c/mL), with phenotypic resistance to INSTI, NNRTI,NRTI and PI were summarized. Assessment of antiviral activity of ART using phenotypic test results was interpreted through a proprietary algorithm (from Monogram Biosciences), which provided the overall susceptibility of the drug. Partially sensitive and resistant calls were considered resistant in this analysis. The phenotypic resistance was calculated using binary scoring system, where 0 was considered as sensitive and 1 as resistance. Phenotypic Resistance data for the following INSTI, NNRTI, NRTI and PI drugs in participants Meeting CVW Criteria has been presented.
Time Frame: Up to Week 48
Population: CVW Population. One participant randomized to TBR but received TDF-based regimen and was presented within the "TBR (TAF-based regimen) arm" as efficacy of TAF and TDF are comparable.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 0 | 1
Participants
  INSTI, DTG, Sensitive |  | 1
  INSTI, DTG, Resistant |  | 0
  INSTI, Bictegravir (BIC), Sensitive |  | 1
  INSTI, BIC, Resistant |  | 0
  INSTI, Elvitegravir (EVG), Sensitive |  | 1
  INSTI, EVG, Resistant |  | 0
  INSTI, Raltegravir (RAL), Sensitive |  | 1
  INSTI, RAL, Resistant |  | 0
  NNRTI, Delavirdine (DLV), Sensitive |  | 1
  NNRTI, DLV, Resistant |  | 0
  NNRTI, Efavirenz (EFV), Sensitive |  | 1
  NNRTI, EFV, Resistant |  | 0
  NNRTI, Etravirine (ETR), Sensitive |  | 1
  NNRTI, ETR, Resistant |  | 0
  NNRTI, Nevirapine (NVP), Sensitive |  | 1
  NNRTI, NVP, Resistant |  | 0
  NNRTI, Rilpivirine (RPV), Sensitive |  | 1
  NNRTI, RPV, Resistant |  | 0
  NRTI, 3TC, Sensitive |  | 1
  NRTI, 3TC, Resistant |  | 0
  NRTI, Abacavir (ABC), Sensitive |  | 1
  NRTI, ABC, Resistant |  | 0
  NRTI, Zidovudine (AZT), Sensitive |  | 1
  NRTI, AZT, Resistant |  | 0
  NRTI, Stavudine (D4T), Sensitive |  | 1
  NRTI, D4T, Resistant |  | 0
  NRTI, Didanosine (DDI), Sensitive |  | 1
  NRTI, DDI, Resistant |  | 0
  NRTI, Emtricitabine (FTC), Sensitive |  | 1
  NRTI, FTC, Resistant |  | 0
  NRTI, Tenofovir (TDF), Sensitive |  | 1
  NRTI, TDF, Resistant |  | 0
  PI, Atazanavir (ATV), Sensitive |  | 1
  PI, ATV, Resistant |  | 0
  PI, Darunavir (DRV), Sensitive |  | 1
  PI, DRV, Resistant |  | 0
  PI, Fosamprenavir (FPV), Sensitive |  | 1
  PI, FPV, Resistant |  | 0
  PI, Indinavir (IDV), Sensitive |  | 1
  PI, IDV, Resistant |  | 0
  PI, Lopinavir (LPV), Sensitive |  | 1
  PI, LPV, Resistant |  | 0
  PI, Nelfinavir (NFV), Sensitive |  | 1
  PI, NFV, Resistant |  | 0
  PI, Ritonavir (RTV), Sensitive |  | 1
  PI, RTV, Resistant |  | 0
  PI, Saquinavir (SQV), Sensitive |  | 1
  PI, SQV, Resistant |  | 0
  PI, Tipranavir (TPV), Sensitive |  | 1
  PI, TPV, Resistant |  | 0

46. Secondary Outcome: Number of Participants With Phenotypic Resistance: Up to Week 144
Description: Number of participants, who meet CVW criteria (one plasma HIV-1 RNA >=200 c/mL after Day 1 with immediate prior HIV RNA >=50 c/mL), with phenotypic resistance to INSTI,NNRT,NRTI and PI were summarized. Assessment of antiviral activity of anti-retroviral therapy (ART) using phenotypic test results was interpreted through a proprietary algorithm (from Monogram Biosciences), which provided the overall susceptibility of the drug. Partially sensitive and resistant calls were considered resistant in this analysis. The phenotypic resistance was calculated using binary scoring system, where 0 was considered as sensitive and 1 as resistance. Phenotypic Resistance data for the following INSTI, NNRTI, NRTI and PI drugs in participants Meeting CVW Criteria has been presented.
Time Frame: Up to Week 144
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 0 | 2
Participants
  INSTI, DTG, Sensitive |  | 2
  INSTI, DTG, Resistant |  | 0
  INSTI, Bictegravir (BIC), Sensitive |  | 2
  INSTI, BIC, Resistant |  | 0
  INSTI, Elvitegravir (EVG), Sensitive |  | 2
  INSTI, EVG, Resistant |  | 0
  INSTI, Raltegravir (RAL), Sensitive |  | 2
  INSTI, RAL, Resistant |  | 0
  NNRTI, Delavirdine (DLV), Sensitive |  | 2
  NNRTI, DLV, Resistant |  | 0
  NNRTI, Efavirenz (EFV), Sensitive |  | 2
  NNRTI, EFV, Resistant |  | 0
  NNRTI, Etravirine (ETR), Sensitive |  | 2
  NNRTI, ETR, Resistant |  | 0
  NNRTI, Nevirapine (NVP), Sensitive |  | 2
  NNRTI, NVP, Resistant |  | 0
  NNRTI, Rilpivirine (RPV), Sensitive |  | 2
  NNRTI, RPV, Resistant |  | 0
  NRTI, 3TC, Sensitive |  | 2
  NRTI, 3TC, Resistant |  | 0
  NRTI, Abacavir (ABC), Sensitive |  | 2
  NRTI, ABC, Resistant |  | 0
  NRTI, Zidovudine (AZT), Sensitive |  | 2
  NRTI, AZT, Resistant |  | 0
  NRTI, Stavudine (D4T), Sensitive |  | 2
  NRTI, D4T, Resistant |  | 0
  NRTI, Didanosine (DDI), Sensitive |  | 2
  NRTI, DDI, Resistant |  | 0
  NRTI, Emtricitabine (FTC), Sensitive |  | 2
  NRTI, FTC, Resistant |  | 0
  NRTI, Tenofovir (TDF), Sensitive |  | 2
  NRTI, TDF, Resistant |  | 0
  PI, Atazanavir (ATV), Sensitive |  | 2
  PI, ATV, Resistant |  | 0
  PI, Darunavir (DRV), Sensitive |  | 2
  PI, DRV, Resistant |  | 0
  PI, Fosamprenavir (FPV), Sensitive |  | 2
  PI, FPV, Resistant |  | 0
  PI, Indinavir (IDV), Sensitive |  | 2
  PI, IDV, Resistant |  | 0
  PI, Lopinavir (LPV), Sensitive |  | 2
  PI, LPV, Resistant |  | 0
  PI, Nelfinavir (NFV), Sensitive |  | 2
  PI, NFV, Resistant |  | 0
  PI, Ritonavir (RTV), Sensitive |  | 2
  PI, RTV, Resistant |  | 0
  PI, Saquinavir (SQV), Sensitive |  | 2
  PI, SQV, Resistant |  | 0
  PI, Tipranavir (TPV), Sensitive |  | 2
  PI, TPV, Resistant |  | 0

47. Secondary Outcome: Change From Baseline in Bone Biomarkers-serum Bone-specific ALP (Bone-ALP), Osteocalcin, Serum Procollagen 1 N-Terminal Propeptide (P1NP) and Serum Type 1 Collagen C-telopeptides (CTX-1) at Weeks 24 and 48
Description: Serum samples were collected for analysis of bone biomarkers. Baseline was latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline is post-dose visit value minus Baseline value. Adjusted mean and its corresponding standard error has been presented. Adjusted mean was the estimated mean change from Baseline at each visit in each arm calculated from a repeated measures model adjusting for treatment, visit, Baseline third agent class, CD4+ cell count (continuous), age (continuous), sex, race, body mass index (BMI) (continuous), smoking status, vitamin D use, Baseline biomarker (continuous), treatment by visit interaction, and Baseline value by visit interaction, with visit as repeated factor.One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 28
Measure: Mean (Standard Error); unit: Micrograms per liter
Groups:
- TAF-based Regimen (Early Switch): Participants who were on a stable TBR and who had an HIV-1 RNA<50 c/mL at the time of screening, were continued to receive TBR up to 48 weeks. One participant randomized to the this arm received TDF rather than TAF-and was presented within the "TAF-based regimen" arm for efficacy because the efficacy of TAF and TDF are comparable. However the participant was presented separately under "TDF-based regimen" for Safety because the safety profiles of TDF and TAF differ.
Arm/Group | DTG+3TC FDC (Early Switch) | TAF-based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Micrograms per liter
  Bone-ALP, Week 24, n=350, 354: number analyzed (Participants) | 350 | 354
  Bone-ALP, Week 24, n=350, 354 | -0.77 (0.112) | -1.05 (0.089)
  Bone-ALP, Week 48, n=343, 342: number analyzed (Participants) | 343 | 342
  Bone-ALP, Week 48, n=343, 342 | -0.03 (0.145) | -0.34 (0.117)
  Osteocalcin, Week 24, n=350 ,353: number analyzed (Participants) | 350 | 353
  Osteocalcin, Week 24, n=350 ,353 | -1.08 (0.248) | 0.26 (0.229)
  Osteocalcin, Week 48, n=343, 342: number analyzed (Participants) | 343 | 342
  Osteocalcin, Week 48, n=343, 342 | -1.15 (0.260) | 0.69 (0.279)
  P1NP, Week24, n=349 ,356: number analyzed (Participants) | 349 | 356
  P1NP, Week24, n=349 ,356 | 7.0 (0.87) | 5.0 (0.72)
  P1NP, Week48, n=342, 343: number analyzed (Participants) | 342 | 343
  P1NP, Week48, n=342, 343 | 9.3 (1.06) | 6.4 (1.00)
  CTX-1, Week 24,n=350,356: number analyzed (Participants) | 350 | 356
  CTX-1, Week 24,n=350,356 | 0.0350 (0.01057) | -0.0031 (0.00833)
  CTX-1, Week 48, n=343, 343: number analyzed (Participants) | 343 | 343
  CTX-1, Week 48, n=343, 343 | 0.0602 (0.01024) | 0.0310 (0.00889)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.047, Mixed Model Repeated Measures; Mean Difference (Net) = 0.29, 95% CI 2-sided [0.00 to 0.57] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for Bone-ALP at Week 24 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.094, Mixed Model Repeated Measures; Mean Difference (Net) = 0.31, 95% CI 2-sided [-0.05 to 0.68] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for Bone-ALP at Week 48 has been presented
Statistical Analysis 3: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -1.34, 95% CI 2-sided [-2.01 to -0.68] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for Osteocalcin at Week 24 has been presented
Statistical Analysis 4: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -1.84, 95% CI 2-sided [-2.59 to -1.09] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for Osteocalcin at Week 48 has been presented
Statistical Analysis 5: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.066, Mixed Model Repeated Measures; Mean Difference (Net) = 2.1, 95% CI 2-sided [-0.1 to 4.3] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for P1NP at Week 24 has been presented
Statistical Analysis 6: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.046, Mixed Model Repeated Measures; Mean Difference (Net) = 2.9, 95% CI 2-sided [0.0 to 5.8] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for P1NP at Week 48 has been presented
Statistical Analysis 7: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.005, Mixed Model Repeated Measures; Mean Difference (Net) = 0.0381, 95% CI 2-sided [0.0117 to 0.0646] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for CTX-1 at Week 24 has been presented
Statistical Analysis 8: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.032, Mixed Model Repeated Measures; Mean Difference (Net) = 0.0292, 95% CI 2-sided [0.0025 to 0.0559] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for CTX-1 at Week 48 has been presented

48. Secondary Outcome: Change From Baseline in Bone Biomarkers-serum Bone-specific ALP (Bone-ALP), Osteocalcin, Serum P1NP and Serum CTX-1 in Participants Randomized to TBR Arm Receiving TDF-based Regimen at Weeks 24 and 48
Description: Serum samples were collected for analysis of bone biomarkers. Baseline was latest pre-dose assessment with a non-missing value (Day 1) . Change from Baseline is post-dose visit value minus Baseline value. Change from Baseline in bone biomarkers-serum bone-specific ALP (Bone-ALP), osteocalcin, serum P1NP and serum CTX-1 in TDF-based regimen participants has been presented. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 29
Measure: Number; unit: Micrograms per liter
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Micrograms per liter
  Bone-ALP, Week 24, n=1 | 0.3
  Bone-ALP, Week 48, n=0: number analyzed (Participants) | 0
  Osteocalcin, Week 24, n=1 | 13.4
  Osteocalcin, Week 48, n=0: number analyzed (Participants) | 0
  P1NP, Week24, n=1 | 11
  P1NP, Week48, n=0: number analyzed (Participants) | 0
  CTX-1, Week 24,n=1 | 0.045
  CTX-1, Week 48, n=0: number analyzed (Participants) | 0

49. Secondary Outcome: Change From Baseline in Bone Biomarkers-serum Bone-ALP, Osteocalcin, Serum P1NP and Serum Type 1 CTX-1 at Weeks 96 and 144
Description: Serum samples were collected for analysis of bone biomarkers. Baseline is latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline is post-dose visit value minus Baseline value. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen"
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: as for outcome 28
Measure: Mean (Standard Error); unit: Micrograms per liter
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Micrograms per liter
  Bone-ALP, Week 96, n=316, 289: number analyzed (Participants) | 316 | 289
  Bone-ALP, Week 96, n=316, 289 | -0.62 (0.145) | -0.79 (0.137)
  Bone-ALP, Week 144, n=314, 301: number analyzed (Participants) | 314 | 301
  Bone-ALP, Week 144, n=314, 301 | -0.27 (0.163) | -0.40 (0.177)
  Osteocalcin, Week 96, n=315 , 288: number analyzed (Participants) | 315 | 288
  Osteocalcin, Week 96, n=315 , 288 | -1.97 (0.288) | -0.10 (0.306)
  Osteocalcin, Week 144, n=315, 301: number analyzed (Participants) | 315 | 301
  Osteocalcin, Week 144, n=315, 301 | -0.74 (0.266) | 1.21 (0.320)
  P1NP, Week 96, n=316 ,290: number analyzed (Participants) | 316 | 290
  P1NP, Week 96, n=316 ,290 | 6.7 (0.87) | 4.7 (0.80)
  P1NP, Week 144, n=315, 302: number analyzed (Participants) | 315 | 302
  P1NP, Week 144, n=315, 302 | 3.9 (0.94) | 3.5 (1.04)
  CTX-1, Week 96 ,n=315, 289: number analyzed (Participants) | 315 | 289
  CTX-1, Week 96 ,n=315, 289 | 0.0201 (0.01123) | 0.0050 (0.00929)
  CTX-1, Week 48, n=315, 300: number analyzed (Participants) | 315 | 300
  CTX-1, Week 48, n=315, 300 | 0.0022 (0.00947) | -0.0104 (0.00907)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.386, Mixed Model Repeated Measures; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.22 to 0.57] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for Bone-ALP at Week 96 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.573, Mixed Model Repeated Measures; Mean Difference (Net) = 0.14, 95% CI 2-sided [-0.34 to 0.61] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for Bone-ALP at Week 144 has been presented
Statistical Analysis 3: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -1.87, 95% CI 2-sided [-2.70 to -1.04] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for Osteocalcin at Week 96 has been presented
Statistical Analysis 4: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -1.95, 95% CI 2-sided [-2.77 to -1.14] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for Osteocalcin at Week 144 has been presented
Statistical Analysis 5: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.082, Mixed Model Repeated Measures; Mean Difference (Net) = 2.1, 95% CI 2-sided [-0.3 to 4.4] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for P1NP at Week 96 has been presented
Statistical Analysis 6: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.765, Mixed Model Repeated Measures; Mean Difference (Net) = 0.4, 95% CI 2-sided [-2.3 to 3.2] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for P1NP at Week 144 has been presented
Statistical Analysis 7: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.301, Mixed Model Repeated Measures; Mean Difference (Net) = 0.0151, 95% CI 2-sided [-0.0136 to 0.0438] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for CTX-1 at Week 96 has been presented
Statistical Analysis 8: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.340, Mixed Model Repeated Measures; Mean Difference (Net) = 0.0126, 95% CI 2-sided [-0.0133 to 0.0384] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for CTX-1 at Week 144 has been presented

50. Secondary Outcome: Change From Baseline in Bone Biomarker: Serum 25-hydroxyvitamin D at Weeks 24 and 48
Description: Serum samples were collected for analysis of 25-hydroxyvitamin D. Baseline value was latest pre-dose assessment (Day 1) with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. Adjusted mean and its corresponding standard error has been presented. Adjusted mean was estimated mean change from Baseline at each visit in each arm calculated from a repeated measures model adjusting for treatment, visit, Baseline third agent class, CD4+ cell count (continuous), age (continuous), sex, race, BMI (continuous), smoking status, vitamin D use, Baseline biomarker (continuous), treatment by visit interaction, and Baseline value by visit interaction, with visit as repeated factor.One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 28
Measure: Mean (Standard Error); unit: Nanomoles per liter
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Nanomoles per liter
  Week 24, n=351, 355: number analyzed (Participants) | 351 | 355
  Week 24, n=351, 355 | 0.0 (1.10) | 2.1 (1.15)
  Week 48, n=344, 343: number analyzed (Participants) | 344 | 343
  Week 48, n=344, 343 | -5.8 (1.21) | -3.5 (1.13)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.173, Mixed Model Repeated Measures; Mean Difference (Net) = -2.2, 95% CI 2-sided [-5.3 to 1.0] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum 25 hydroxyvitamin D at Week 24 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.168, Mixed Model Repeated Measures; Mean Difference (Net) = -2.3, 95% CI 2-sided [-5.5 to 1.0] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum 25 hydroxyvitamin D at Week 48 has been presented

51. Secondary Outcome: Change From Baseline in Bone Biomarker: Serum 25-hydroxyvitamin D at Weeks 24 and 48 in Participants Randomized to TBR Arm Receiving TDF-based Regimen
Description: Serum samples were collected for the analysis of 25-hydroxyvitamin D. Baseline value was the value from latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. Change from Baseline values for serum 25-hydroxyvitamin D in TDF-based regimen participants has been presented. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 29
Measure: Number; unit: Nanomoles per liter
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Nanomoles per liter
  Week 24, n=1 | 2
  Week 48, n=0: number analyzed (Participants) | 0

52. Secondary Outcome: Change From Baseline in Bone Biomarker: Serum 25-hydroxyvitamin D at Weeks 96 and 144
Description: Serum samples were collected for analysis of 25-hydroxyvitamin D. Baseline value is latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen"
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: as for outcome 28
Measure: Mean (Standard Error); unit: Nanomoles per liter
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Nanomoles per liter
  Week 96, n=315, 291: number analyzed (Participants) | 315 | 291
  Week 96, n=315, 291 | -11.5 (1.17) | -2.2 (2.06)
  Week 144, n=315, 303: number analyzed (Participants) | 315 | 303
  Week 144, n=315, 303 | -7.5 (1.28) | -1.9 (1.50)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -9.4, 95% CI 2-sided [-14.0 to -4.7] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum 25 hydroxyvitamin D at Week 96 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.005, Mixed Model Repeated Measures; Mean Difference (Net) = -5.6, 95% CI 2-sided [-9.4 to -1.7] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum 25 hydroxyvitamin D at Week 144 has been presented

53. Secondary Outcome: Change From Baseline in Renal Biomarker- Serum Cystatin C at Weeks 24 and 48
Description: Serum samples were collected to assess renal biomarker. Baseline was latest pre-dose assessment value with non-missing value (Day 1). Change from Baseline is post-dose visit value minus Baseline value. Adjusted mean and its corresponding standard error has been presented. Adjusted mean was estimated mean change from Baseline at each visit in each arm calculated from a repeated measures model adjusting for following:treatment, visit, Baseline third agent class, CD4+ cell count(continuous), age(continuous), sex, race, BMI(continuous), presence of diabetes mellitus, presence of hypertension, Baseline biomarker(continuous), treatment by visit interaction, and Baseline value by visit interaction, with visit as repeated factor. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen"
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 28
Measure: Mean (Standard Error); unit: Milligrams per liter
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Milligrams per liter
  Week 24, n=351, 357: number analyzed (Participants) | 351 | 357
  Week 24, n=351, 357 | -0.03 (0.005) | -0.02 (0.004)
  Week 48, n=344, 343: number analyzed (Participants) | 344 | 343
  Week 48, n=344, 343 | 0.00 (0.006) | 0.01 (0.005)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.027, Mixed Model Repeated Measures; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.03 to 0.00] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum cystatin C at Week 24 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.061, Mixed Model Repeated Measures; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.03 to 0.00] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum cystatin C at Week 48 has been presented

54. Secondary Outcome: Change From Baseline in Renal Biomarker- Serum Cystatin C at Weeks 24 and 48 in Participants Randomized to TBR Arm Receiving TDF-based Regimen
Description: Serum samples were collected at Baseline, Week 24 and Week 48 to assess renal inflammation biomarker - cystatin C. Baseline was defined as the latest pre-dose assessment value with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. Change from Baseline values for serum cystatin -C biomarker in TDF based regimen participants has been presented. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 29
Measure: Number; unit: Milligrams per liter
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Milligrams per liter
  Week 24, n=1 | 0
  Week 48, n=0: number analyzed (Participants) | 0

55. Secondary Outcome: Change From Baseline in Renal Biomarker- Serum Cystatin C at Weeks 96 and 144
Description: Serum samples were collected to assess renal biomarker. Baseline is latest pre-dose assessment value with non-missing value (Day 1). Change from Baseline is post-dose visit value minus Baseline value. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen"
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: as for outcome 28
Measure: Mean (Standard Error); unit: Milligrams per liter
Arm/Group | DTG+3TC FDC (Early Switch) | TAF-based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Milligrams per liter
  Week 96, n=316, 290: number analyzed (Participants) | 316 | 290
  Week 96, n=316, 290 | 0.07 (0.008) | 0.10 (0.009)
  Week 144, n=315, 302: number analyzed (Participants) | 315 | 302
  Week 144, n=315, 302 | 0.13 (0.006) | 0.14 (0.006)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.004, Mixed Model Repeated Measures; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.06 to -0.01] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum cystatin C at Week 96 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p = 0.094, Mixed Model Repeated Measures; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.03 to 0.00] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum cystatin C at Week 144 has been presented

56. Secondary Outcome: Change From Baseline in Renal Biomarker- Serum GFR From Cystatin C Adjusted Using CKD-EPI and Serum GFR From Creatinine Adjusted Using CKD-EPI at Weeks 24 and 48
Description: Serum samples assessed:serum GFR from cystatin C and from creatinine adjusted using CKD-EPI Baseline(Day 1) was value from latest pre-dose assessment with non-missing value. Change from Baseline is post-dose visit value minus Baseline value.Adjusted mean and standard error is presented.Adjusted mean was estimated mean change from Baseline at each visit in each arm calculated from repeated measures model adjusting for treatment, visit, Baseline third agent class,CD4+ cell count(continuous),age(continuous), sex, race, BMI(continuous),presence of diabetes mellitus, presence of hypertension, Baseline biomarker(continuous), treatment by visit interaction, and Baseline value by visit interaction, with visit as repeated factor. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen"
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 28
Measure: Mean (Standard Error); unit: Milliliters/minute/1.73*meter square
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Milliliters/minute/1.73*meter square
  GFR from cystatin C CKD-EPI, Week 24, n=351, 357: number analyzed (Participants) | 351 | 357
  GFR from cystatin C CKD-EPI, Week 24, n=351, 357 | 3.2 (0.52) | 1.5 (0.46)
  GFR from cystatin C CKD-EPI, Week 48, n=344, 343: number analyzed (Participants) | 344 | 343
  GFR from cystatin C CKD-EPI, Week 48, n=344, 343 | 0.1 (0.61) | -1.6 (0.59)
  GFR from creatinine CKD-EPI, Week 24, n=351, 359: number analyzed (Participants) | 351 | 359
  GFR from creatinine CKD-EPI, Week 24, n=351, 359 | -8.8 (0.48) | -3.8 (0.47)
  GFR from creatinine CKD-EPI, Week 48, n=344, 345: number analyzed (Participants) | 344 | 345
  GFR from creatinine CKD-EPI, Week 48, n=344, 345 | -7.7 (0.48) | -2.9 (0.48)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.012, Mixed Model Repeated Measures; Mean Difference (Net) = 1.8, 95% CI 2-sided [0.4 to 3.1] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum GFR from cystatin C adjusted using CKD-EPI at Week 24 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.059, Mixed Model Repeated Measures; Mean Difference (Net) = 1.6, 95% CI 2-sided [-0.1 to 3.3] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum GFR from cystatin C adjusted using CKD-EPI at Week 48 has been presented
Statistical Analysis 3: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -5.0, 95% CI 2-sided [-6.3 to -3.7] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum GFR from creatinine adjusted using CKD-EPI at Week 24 has been presented
Statistical Analysis 4: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -4.8, 95% CI 2-sided [-6.1 to -3.4] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum GFR from creatinine adjusted using CKD-EPI at Week 48 has been presented

57. Secondary Outcome: Change From Baseline in Renal Biomarker- Serum GFR From Cystatin C Adjusted Using CKD-EPI and Serum GFR From Creatinine Adjusted Using CKD-EPI at Weeks 24 and 48 in Participants Randomized to TBR Arm Receiving TDF-based Regimen
Description: Serum samples were collected at Baseline, Week 24 and Week 48 to assess renal inflammation biomarkers - serum GFR from cystatin C adjusted using CKD-EPI and serum GFR from creatinine adjusted using CKD-EPI. Baseline was defined as the latest pre-dose assessment value with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. Change from Baseline in serum GFR from cystatin C adjusted using CKD-EPI and serum GFR from creatinine adjusted using CKD-EPI in TDF-based regimen participants has been presented. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 29
Measure: Number; unit: Milliliters/minute/1.73*meter square
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Milliliters/minute/1.73*meter square
  GFR from cystatin C CKD-EPI, Week 24, n=1 | 0
  GFR from cystatin C CKD-EPI, Week 48, n=0: number analyzed (Participants) | 0
  GFR from creatinine CKD-EPI, Week 24, n=1 | 4
  GFR from creatinine CKD-EPI, Week 48, n=0: number analyzed (Participants) | 0

58. Secondary Outcome: Change From Baseline in Renal Biomarker- Serum GFR From Cystatin C Adjusted Using CKD-EPI and Serum GFR From Creatinine Adjusted Using CKD-EPI at Weeks 96 and 144
Description: Serum samples were collected to assess serum GFR from cystatin C and from creatinine adjusted for BSA. Baseline is defined as the latest pre-dose assessment value with a non-missing value (Day 1). Change from Baseline is post-dose visit value minus Baseline value. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen"
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: as for outcome 28
Measure: Mean (Standard Error); unit: Milliliters/minute/1.73*meter square
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Milliliters/minute/1.73*meter square
  GFR from cystatin C CKD-EPI, Week 96, n=316, 290: number analyzed (Participants) | 316 | 290
  GFR from cystatin C CKD-EPI, Week 96, n=316, 290 | -7.6 (0.89) | -11.7 (0.99)
  GFR from cystatin C CKD-EPI, Week 144, n=315, 302: number analyzed (Participants) | 315 | 302
  GFR from cystatin C CKD-EPI, Week 144, n=315, 302 | -13.9 (0.71) | -15.8 (0.70)
  GFR from creatinine adjusted for BSA, Week 96, n=315, 294: number analyzed (Participants) | 315 | 294
  GFR from creatinine adjusted for BSA, Week 96, n=315, 294 | -7.2 (0.55) | -1.9 (0.52)
  GFR from creatinine adjusted for BSA, Week 144, n=311, 300: number analyzed (Participants) | 311 | 300
  GFR from creatinine adjusted for BSA, Week 144, n=311, 300 | -11.5 (0.62) | -7.0 (0.60)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.002, Mixed Model Repeated Measures; Mean Difference (Net) = 4.1, 95% CI 2-sided [1.5 to 6.7] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum GFR from cystatin C adjusted using CKD-EPI at Week 96 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.064, Mixed Model Repeated Measures; Mean Difference (Net) = 1.9, 95% CI 2-sided [-0.1 to 3.8] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum GFR from cystatin C adjusted using CKD-EPI at Week 148 has been presented
Statistical Analysis 3: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -5.2, 95% CI 2-sided [-6.7 to -3.8] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum GFR from creatinine adjusted using CKD-EPI at Week 96 has been presented
Statistical Analysis 4: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -4.5, 95% CI 2-sided [-6.2 to -2.8] — Mean difference (DTG+3TC - TAF based regimen) and its 95% CI for serum GFR from creatinine adjusted using CKD-EPI at Week 144 has been presented

59. Secondary Outcome: Change From Baseline in Renal Biomarker- Serum Creatinine at Weeks 24 and 48
Description: Serum samples assessed: renal inflammation biomarker serum creatinine.Baseline(Day 1)was value from latest pre-dose assessment with non-missing value. Change from Baseline is post-dose visit value minus Baseline value. Adjusted mean and its corresponding standard error has been presented. Adjusted mean was estimated mean change from Baseline at each visit in each arm calculated from repeated measures model adjusting for treatment, visit, Baseline third agent class, CD4+ cell count(continuous), age(continuous), sex, race, BMI(continuous), presence of diabetes mellitus, presence of hypertension, Baseline biomarker(continuous), treatment by visit interaction, Baseline value by visit interaction, with visit as repeated factor. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen"
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 28
Measure: Mean (Standard Error); unit: Micromoles per liter
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Micromoles per liter
  Week 24, n=351, 359: number analyzed (Participants) | 351 | 359
  Week 24, n=351, 359 | 7.47 (0.466) | 3.11 (0.495)
  Week 48, n=344, 345: number analyzed (Participants) | 344 | 345
  Week 48, n=344, 345 | 6.67 (0.493) | 2.18 (0.450)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = 4.37, 95% CI 2-sided [3.03 to 5.70] — Mean difference (DTG+3TC - TBR) and its 95% CI for serum creatinine at Week 24 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = 4.49, 95% CI 2-sided [3.18 to 5.81] — Mean difference (DTG+3TC - TBR) and its 95% CI for serum creatinine at Week 48 has been presented

60. Secondary Outcome: Change From Baseline in Renal Biomarker- Serum Creatinine at Weeks 24 and 48 in Participants Randomized to TBR Arm Receiving TDF-based Regimen
Description: Serum samples were collected at Baseline, Week 24 and Week 48 to assess renal inflammation biomarker - serum creatinine. Baseline was defined as the latest pre-dose assessment value with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value. Change from Baseline in serum creatinine in TDF-based regimen participants has been presented. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen."
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 29
Measure: Number; unit: Micromoles per liter
Arm/Group | Randomized to TBR But Received TDF-based Regimen (Early Switch)
Number analyzed (Participants) | 1
Micromoles per liter
  Week 24, n=1 | -8
  Week 48, n=0: number analyzed (Participants) | 0

61. Secondary Outcome: Change From Baseline in Renal Biomarker- Serum Creatinine at Weeks 96 and 144
Description: Serum samples were collected to assess renal inflammation biomarker - serum creatinine. Baseline is defined as the latest pre-dose assessment value with a non-missing value (Day 1). Change from Baseline is post-dose visit value minus Baseline value. One participant randomized to TBR but received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen"
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: Safety Population. Total of 741 participants were analyzed but 740 participants are presented in this Outcome Measure and 1 participant is presented separately in next Outcome Measure. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Error); unit: Micromoles per liter
Arm/Group | DTG+3TC FDC (Early Switch) | TAF-based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 371
Micromoles per liter
  Week 96, n=316, 294: number analyzed (Participants) | 316 | 294
  Week 96, n=316, 294 | 5.53 (0.553) | 0.58 (0.515)
  Week 144, n=311, 302: number analyzed (Participants) | 311 | 302
  Week 144, n=311, 302 | 9.25 (0.637) | 5.17 (0.633)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = 4.95, 95% CI 2-sided [3.47 to 6.43] — Mean difference (DTG+3TC - TBR) and its 95% CI for serum creatinine at Week 96 has been presented
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF-based Regimen (Early Switch); Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = 4.08, 95% CI 2-sided [2.32 to 5.85] — Mean difference (DTG+3TC - TBR) and its 95% CI for serum creatinine at Week 144 has been presented

62. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Utility Score at Week 24 and 48
Description: EQ-5D-5L questionnaire provides a profile of participant function and a global health state rating. The five-item measure has one question assessing each of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 5 levels for each dimension including 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. The health state is defined by combining the levels of answers from each of the 5 questions. Each health state is referred to in terms of a 5 digit code. Health state 5 digit code is translated into utility score, which is valued up to 1 (perfect health) with lower values meaning worse state. EQ-5D-5L utility score ranges from -0.281 to 1. Higher scores indicate better health.
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: ITT-E Population. One participant randomized to TBR but received TDF-based regimen and was presented within the "TBR (TAF-based regimen) arm" as efficacy of TAF and TDF are comparable. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 364 | 370
Scores on a scale
  Week 24 | 0.0029 (0.00383) | 0.0046 (0.00352)
  Week 48 | 0.0037 (0.00407) | 0.0023 (0.00373)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.741, Mixed Model Repeated Measures; Mean Difference (Net) = -0.0017, 95% CI 2-sided [-0.0119 to 0.0085] — Week 24. MMRM adjusted for following: Treatment, Visit, Baseline Third Agent Class, Baseline EQ-5D Utility (continuous), Treatment by Visit interaction, and Baseline EQ-5D Utility by Visit interaction, with Visit as the repeated factor
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.792, Mixed Model Repeated Measures; Mean Difference (Net) = 0.0015, 95% CI 2-sided [-0.0094 to 0.0123] — Week 48. MMRM adjusted for following: Treatment, Visit, Baseline Third Agent Class, Baseline EQ-5D Utility (continuous), Treatment by Visit interaction, and Baseline EQ-5D Utility by Visit interaction, with Visit as the repeated factor

63. Secondary Outcome: Change From Baseline in EQ-5D-5L Utility Score at Weeks 96 and 144
Description: EQ-5D-5L questionnaire provides profile of participant function and global health state rating. Five-item measure has 1question assessing each of 5dimensions:mobility,self-care,usual activities,pain/discomfort,anxiety/depression and 5 levels for each dimension including 1=no problems,2=slight problems,3=moderate problems,4=severe problems,5=extreme problems. Health state is defined by combining levels of answers from each of 5 questions. Each health state is referred to in terms of a 5 digit code.Health state 5 digit code is translated into utility score, which is valued up to 1 (perfect health) with lower values meaning worse state.EQ-5D-5L utility score ranges from -0.281 to 1. Higher scores indicate better health.Baseline is latest pre-dose assessment value with a non-missing value (Day 1).Change from Baseline is post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: ITT-E Population. One participant randomized to TBR but received TDF-based regimen and was presented within the "TBR (TAF-based regimen) arm" as efficacy of TAF and TDF are comparable. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 372
Scores on a scale
  Week 96, n=364, 370: number analyzed (Participants) | 364 | 370
  Week 96, n=364, 370 | -0.0036 (0.00442) | -0.0038 (0.00446)
  Week 144, n=364, 369: number analyzed (Participants) | 364 | 369
  Week 144, n=364, 369 | -0.0151 (0.00502) | -0.0042 (0.00492)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.965, Mixed Model Repeated Measures; Mean Difference (Net) = 0.0003, 95% CI 2-sided [-0.0121 to 0.0126] — Week 96. MMRM adjusted for following: Treatment, Visit, Baseline Third Agent Class, Baseline EQ-5D Utility (continuous), Treatment by Visit interaction, and Baseline EQ-5D Utility by Visit interaction, with Visit as the repeated factor
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.120, Mixed Model Repeated Measures; Mean Difference (Net) = -0.0109, 95% CI 2-sided [-0.0247 to 0.0029] — Week 144. MMRM adjusted for following: Treatment, Visit, Baseline Third Agent Class, Baseline EQ-5D Utility (continuous), Treatment by Visit interaction, and Baseline EQ-5D Utility by Visit interaction, with Visit as the repeated factor

64. Secondary Outcome: Change From Baseline in EQ-5D-5L Thermometer Scores at Week 24 and 48
Description: EQ-5D-5L questionnaire provides a profile of participant function and a global health state rating. The five-item measure has one question assessing each of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 5 levels for each dimension including 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. EQ-5D-5L included EQ visual Analogue scale (EQ VAS) 'Thermometer' which provided Self-rated current health status. Score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). MMRM was run on the LOCF dataset. Baseline was the latest pre-dose assessment value with a non-missing value (Day 1) and change from Baseline is defined as post-dose value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 62
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 364 | 369
Scores on a scale
  Week 24 | 1.2 (0.49) | 1.3 (0.44)
  Week 48 | 1.1 (0.52) | 1.7 (0.43)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.879, Mixed Model Repeated Measures; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.4 to 1.2] — Week 24. MMRM adjusted for following: Treatment, Visit, Baseline Third Agent Class, Baseline EQ-5D Thermometer (continuous), Treatment by Visit interaction, and Baseline EQ-5D Thermometer by Visit interaction, with Visit as the repeated factor
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.414, Mixed Model Repeated Measures; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.9 to 0.8] — Week 48. MMRM adjusted for following: Treatment, Visit, Baseline Third Agent Class, Baseline EQ-5D Thermometer (continuous), Treatment by Visit interaction, and Baseline EQ-5D Thermometer by Visit interaction, with Visit as the repeated factor

65. Secondary Outcome: Change From Baseline in EQ-5D-5L Thermometer Scores at Weeks 96 and 144
Description: EQ-5D-5L questionnaire provides a profile of participant function and a global health state rating. The five-item measure has one question assessing each of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 5 levels for each dimension including 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. EQ-5D-5L included EQ visual Analogue scale (EQ VAS) 'Thermometer' which provided Self-rated current health status. Score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). Baseline is defined as the latest pre-dose assessment value with a non-missing value (Day 1). Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 96 and 144
Population: as for outcome 63
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG+3TC FDC (Early Switch) | TAF Based Regimen (Early Switch)
Number analyzed (Participants) | 369 | 372
Scores on a scale
  Week 96, n=364, 369: number analyzed (Participants) | 364 | 369
  Week 96, n=364, 369 | 0.7 (0.52) | 1.9 (0.48)
  Week 144, n=364, 368: number analyzed (Participants) | 364 | 368
  Week 144, n=364, 368 | 0.2 (0.58) | 1.4 (0.50)
Statistical Analysis 1: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.102, Mixed Model Repeated Measures; Mean Difference (Net) = -1.2, 95% CI 2-sided [-2.5 to 0.2] — Week 96. MMRM adjusted for following: Treatment, Visit, Baseline Third Agent Class, Baseline EQ-5D Thermometer (continuous), Treatment by Visit interaction, and Baseline EQ-5D Thermometer by Visit interaction, with Visit as the repeated factor
Statistical Analysis 2: Comparison: DTG+3TC FDC (Early Switch) vs TAF Based Regimen (Early Switch); Test type: Other; p = 0.093, Mixed Model Repeated Measures; Mean Difference (Net) = -1.3, 95% CI 2-sided [-2.8 to 0.2] — Week 144. MMRM adjusted for following: Treatment, Visit, Baseline Third Agent Class, Baseline EQ-5D Thermometer (continuous), Treatment by Visit interaction, and Baseline EQ-5D Thermometer by Visit interaction, with Visit as the repeated factor

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-serious AEs were collected for DTG + 3TC FDC (Early Switch + Late Switch)-Overall arm up to Week 196; TAF Based Regimen (Early Switch) up to Week 148; for Randomized to TBR but received TDF-based regimen arm up to week 48; and for TAF Based Regimen (Early Switch) followed by DTG + 3TC FDC (Late Switch) from Week 148 to Week 196
Description: Safety Population. One participant randomized to TBR received TDF-based regimen and because the safety profiles of TDF and TAF differ, this participant was removed from the overall safety population and is presented in separate arm "Randomized to TBR but received TDF-based regimen (Early switch)". Data was not collected for "Randomized to TBR But Received TDF-based Regimen (Early switch)" arm at Week 148 as the participant withdrew from the study at Week 36
Groups:
- DTG + 3TC FDC (Early Switch + Late Switch)-Overall: Participants who were on a stable TBR and who had an HIV-1 ribonucleic acid (RNA) <50 copies per millilter (c/mL) at the time of screening, received fixed dose combination of DTG 50 mg + 3TC 300 mg once daily up to 196 weeks during early and late switch phase.
- TAF Based Regimen (Early Switch): Participants who were on a stable TBR and who had an HIV-1 RNA<50 c/mL at the time of screening, were continued to receive TBR up to 148 weeks during early switch phase.
- TAF Based Regimen (Early Switch) Followed by DTG + 3TC FDC (Late Switch): Participants who were on a stable TBR and who had an HIV-1 RNA<50 c/mL at the time of screening, were continued to receive TBR up to 148 weeks during early switch phase. At Week 148 (or upon retest) were switched to DTG/3TC FDC once daily up to Week 196 during late switch phase.
Arm/Group | DTG + 3TC FDC (Early Switch + Late Switch)-Overall | TAF Based Regimen (Early Switch) | Randomized to TBR But Received TDF-based Regimen (Early Switch) | TAF Based Regimen (Early Switch) Followed by DTG + 3TC FDC (Late Switch)
All-Cause Mortality (participants affected / at risk) | 4/369 | 0/371 | 0/1 | 0/298
Serious Adverse Events (participants affected / at risk) | 65/369 | 44/371 | 0/1 | 15/298
Other Adverse Events (participants affected / at risk) | 327/369 | 304/371 | 1/1 | 187/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG + 3TC FDC (Early Switch + Late Switch)-Overall (N=369) | TAF Based Regimen (Early Switch) (N=371) | Randomized to TBR But Received TDF-based Regimen (Early Switch) (N=1) | TAF Based Regimen (Early Switch) Followed by DTG + 3TC FDC (Late Switch) (N=298)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amniotic cavity infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Meningitis pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shigella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthritis gonococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis intestinal perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Bipolar II disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Burkitt's lymphoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiplegic migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nose deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sacroiliac joint dysfunction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type I hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG + 3TC FDC (Early Switch + Late Switch)-Overall (N=369) | TAF Based Regimen (Early Switch) (N=371) | Randomized to TBR But Received TDF-based Regimen (Early Switch) (N=1) | TAF Based Regimen (Early Switch) Followed by DTG + 3TC FDC (Late Switch) (N=298)
Nasopharyngitis (Infections and infestations) | 71 (109) | 64 (93) | 0 (0) | 16 (18)
Upper respiratory tract infection (Infections and infestations) | 52 (72) | 42 (56) | 1 (1) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 54 (70) | 43 (55) | 1 (1) | 12 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 47 (53) | 49 (63) | 0 (0) | 11 (12)
Headache (Nervous system disorders) | 41 (54) | 23 (33) | 0 (0) | 17 (20)
Syphilis (Infections and infestations) | 49 (61) | 33 (43) | 0 (0) | 13 (13)
Gastroenteritis (Infections and infestations) | 29 (37) | 23 (26) | 0 (0) | 5 (5)
Bronchitis (Infections and infestations) | 17 (19) | 23 (24) | 0 (0) | 5 (5)
Anxiety (Psychiatric disorders) | 43 (44) | 29 (30) | 0 (0) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 (56) | 39 (43) | 0 (0) | 15 (17)
Pharyngitis (Infections and infestations) | 21 (22) | 22 (25) | 0 (0) | 5 (5)
Vitamin D deficiency (Metabolism and nutrition disorders) | 22 (23) | 12 (15) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 23 (25) | 18 (20) | 0 (0) | 4 (4)
Anal chlamydia infection (Infections and infestations) | 13 (16) | 22 (31) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 31 (32) | 21 (24) | 0 (0) | 6 (6)
Influenza (Infections and infestations) | 18 (18) | 14 (14) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 29 (34) | 18 (18) | 0 (0) | 7 (8)
Abdominal pain (Gastrointestinal disorders) | 19 (21) | 14 (15) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 15 (15) | 11 (11) | 0 (0) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (30) | 20 (21) | 0 (0) | 5 (5)
Seasonal allergy (Immune system disorders) | 15 (18) | 4 (5) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 16 (19) | 12 (14) | 0 (0) | 3 (4)
Toothache (Gastrointestinal disorders) | 13 (15) | 16 (19) | 0 (0) | 4 (5)
Urethritis (Infections and infestations) | 16 (21) | 13 (14) | 0 (0) | 5 (5)
Erectile dysfunction (Reproductive system and breast disorders) | 15 (15) | 19 (20) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 (25) | 14 (17) | 0 (0) | 6 (7)
Vomiting (Gastrointestinal disorders) | 12 (12) | 6 (6) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 10 (12) | 12 (12) | 0 (0) | 0 (0)
Proctitis gonococcal (Infections and infestations) | 15 (20) | 11 (15) | 0 (0) | 4 (5)
Constipation (Gastrointestinal disorders) | 15 (19) | 7 (7) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 76 (79) | 25 (25) | 0 (0) | 55 (57)
Chlamydial infection (Infections and infestations) | 21 (23) | 12 (12) | 0 (0) | 6 (6)
Oropharyngeal gonococcal infection (Infections and infestations) | 16 (22) | 15 (16) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 13 (15) | 15 (17) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 16 (19) | 8 (10) | 0 (0) | 2 (2)
Folliculitis (Infections and infestations) | 0 (0) | 14 (16) | 0 (0) | 0 (0)
Gonorrhoea (Infections and infestations) | 12 (15) | 9 (10) | 0 (0) | 5 (7)
Tonsillitis (Infections and infestations) | 8 (13) | 10 (12) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 9 (11) | 9 (9) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 10 (13) | 10 (12) | 0 (0) | 7 (8)
Urethritis gonococcal (Infections and infestations) | 15 (16) | 4 (4) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 10 (11) | 6 (7) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 9 (9) | 2 (2) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 8 (10) | 11 (13) | 0 (0) | 0 (0)
Proctitis chlamydial (Infections and infestations) | 14 (23) | 0 (0) | 0 (0) | 2 (2)
Suspected COVID-19 (Infections and infestations) | 8 (9) | 0 (0) | 0 (0) | 2 (2)
Tinea versicolour (Infections and infestations) | 8 (11) | 0 (0) | 0 (0) | 1 (1)
Urethritis chlamydial (Infections and infestations) | 8 (11) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 20 (20) | 9 (12) | 0 (0) | 6 (6)
Haemorrhoids (Gastrointestinal disorders) | 14 (14) | 12 (12) | 0 (0) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 11 (13) | 9 (9) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 5 (5) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 10 (11) | 6 (6) | 0 (0) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 9 (9) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 8 (9) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 9 (9) | 0 (0) | 0 (0) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (10) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 6 (6) | 0 (0) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 0 (0) | 0 (0) | 4 (4)
Migraine (Nervous system disorders) | 9 (10) | 5 (5) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 17 (17) | 0 (0) | 2 (2)
Fatigue (General disorders) | 32 (33) | 11 (12) | 0 (0) | 11 (11)
Pyrexia (General disorders) | 19 (20) | 14 (15) | 0 (0) | 7 (8)
Influenza like illness (General disorders) | 0 (0) | 13 (16) | 0 (0) | 0 (0)
Chest pain (General disorders) | 9 (10) | 9 (10) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11) | 12 (13) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 15 (17) | 11 (11) | 0 (0) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 10 (10) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (9) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 8 (12) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 8 (9) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 8 (8) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 8 (9) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 8 (8) | 0 (0) | 0 (0) | 5 (5)
Muscle strain (Injury, poisoning and procedural complications) | 8 (8) | 4 (4) | 0 (0) | 1 (1)
Weight increased (Investigations) | 9 (9) | 19 (19) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 26 (28) | 15 (15) | 0 (0) | 7 (7)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (10) | 10 (11) | 0 (0) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 8 (8) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 8 (8) | 0 (0) | 0 (0) | 3 (3)
Dysuria (Renal and urinary disorders) | 9 (9) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 8 (8) | 0 (0) | 0 (0) | 2 (2)
Abnormal weight gain (Metabolism and nutrition disorders) | 12 (12) | 0 (0) | 0 (0) | 4 (4)
Abnormal loss of weight (Metabolism and nutrition disorders) | 10 (10) | 0 (0) | 0 (0) | 1 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 (9) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 (9) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT03446573/Prot_002.pdf
  • Statistical Analysis Plan (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT03446573/SAP_003.pdf